CLINICAL TRIAL: NCT01190202
Title: Epidemiology Study of Malaria Transmission Intensity in Sub-Saharan Africa
Brief Title: Epidemiology Study of Malaria Transmission Intensity in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: 114001
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Blood Specimen Collection

ARMS (4):
- Overall Study Group (Survey 1) (Experimental): Subjects at least 6 months of age at the time of Survey 1, conducted at Year 1 of the 4 annual cross sectional surveys performed preferably at peak transmission (end of rainy season), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy. Subjects were enrolled from the catchment areas of study 110021 (NCT00866619) but those who previously participated in study 110021 were excluded from this epidemiological study.
  Interventions: Procedure: Blood sampling; Procedure: Assessment of body temperature
- Overall Study Group (Survey 2) (Experimental): Subjects at least 6 months of age at the time of Survey 2, conducted at Year 2 of the 4 annual cross sectional surveys performed preferably at peak transmission (end of rainy season), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy. Subjects were enrolled from the catchment areas of study 110021 (NCT00866619) but those who previously participated in study 110021 were excluded from this epidemiological study.
  Interventions: Procedure: Blood sampling; Procedure: Assessment of body temperature
- Overall Study Group (Survey 3) (Experimental): Subjects at least 6 months of age at the time of Survey 3, conducted at Year 3 of the 4 annual cross sectional surveys performed preferably at peak transmission (end of rainy season), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy. Subjects were enrolled from the catchment areas of study 110021 (NCT00866619) but those who previously participated in study 110021 were excluded from this epidemiological study.
  Interventions: Procedure: Blood sampling; Procedure: Assessment of body temperature
- Overall Study Group (Survey 4) (Experimental): Subjects at least 6 months of age at the time of Survey 4, conducted at Year 4 of the 4 annual cross sectional surveys performed preferably at peak transmission (end of rainy season), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy. Subjects were enrolled from the catchment areas of study 110021 (NCT00866619) but those who previously participated in study 110021 were excluded from this epidemiological study.
  Interventions: Procedure: Blood sampling; Procedure: Assessment of body temperature

INTERVENTIONS:
Procedure: Blood sampling — Capillary blood samples collected by finger/heel prick
Procedure: Assessment of body temperature — Assessment of axial body temperature with a digital thermometer

SUMMARY:
The aim of this epidemiology study is to characterize in a standardized way malaria transmission intensity at the clinical trial centers participating in study 110021 (NCT00866619).

DETAILED DESCRIPTION:
This study is a multicenter epidemiology study at centers that are participating in GSK's pivotal Phase III candidate malaria vaccine 110021 ( NCT00866619) trial and will involve 4 annual cross sectional surveys performed preferably at peak transmission.

There will be no study vaccine administered in this epidemiology study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female 6 months or older at the time of survey.
* Written informed consent obtained from the subject/from the parent(s)/ Legally Acceptable Representative(s) of the subject.

Exclusion Criteria:

* Child in care.
* Previous or current participation in any malaria vaccine trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21618 (Actual)
Dates: Start 2011-03-14 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2013-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- GSK Investigational Site, Ouagadougou, Burkina Faso
- GSK Investigational Site, Lambaréné, Gabon
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Kumasi
- GSK Investigational Site, Kisumu, Kenya
- GSK Investigational Site, Lilongwe, Malawi
- Tanzania (2):
  - GSK Investigational Site, Dar es Salaam
  - GSK Investigational Site, Korogwe, Tanga

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=5123

REFERENCES:
- [Background] Drakeley C, Abdulla S, Agnandji ST, Fernandes JF, Kremsner P, Lell B, Mewono L, Bache BE, Mihayo MG, Juma O, Tanner M, Tahita MC, Tinto H, Diallo S, Lompo P, D'Alessandro U, Ogutu B, Otieno L, Otieno S, Otieno W, Oyieko J, Asante KP, Dery DB, Adjei G, Adeniji E, Atibilla D, Owusu-Agyei S, Greenwood B, Gesase S, Lusingu J, Mahende C, Mongi R, Segeja M, Adjei S, Agbenyega T, Agyekum A, Ansong D, Bawa JT, Boateng HO, Dandalo L, Escamilla V, Hoffman I, Maenje P, Martinson F, Carter T, Leboulleux D, Kaslow DC, Usuf E, Pircon JY, Bahmanyar ER. Longitudinal estimation of Plasmodium falciparum prevalence in relation to malaria prevention measures in six sub-Saharan African countries. Malar J. 2017 Oct 27;16(1):433. doi: 10.1186/s12936-017-2078-3. PMID 29078773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For each year and each site, approximately 400 subjects at least 6 months and < 5 years old, approximately 200 subjects at least 5 years and < 20 years old and approximately 200 subjects at least 20 years old were to be enrolled. The study was conducted at 8 sites and 6 countries for the first 3 surveys and 3 sites from 3 countries for Survey 4.
Period: Overall Study
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Started | 6404 | 6414 | 6400 | 2400
Completed | 6404 | 6414 | 6400 | 2400
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4) | Total
Number analyzed (Participants) | 6404 | 6414 | 6400 | 2400 | 21618
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.6 (14.6) | 12.1 (14.3) | 12.1 (14.2) | 12.4 (14.4) | 12.28 (14.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3670 | 3791 | 3752 | 1420 | 12633
  Male | 2734 | 2623 | 2648 | 980 | 8985
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasmodium Falciparum (P. Falciparum) Parasitaemia (PFP), for Each Survey
Description: The Overall parasite prevalence (PP) data were collected across centers from subjects aged between and including: 6 months to 4 Years (6M-4Y), 5 to 19 Years (5-19 Y) and 20 Years or older (20Y+), for each Survey. The number of subjects P. Falciparum parasitemia infected among the number of subjects with known result for P.falciparum parasitemia test was tabulated.
Time Frame: At each Survey visit
Population: Analysis was performed on the According-to-Protocol (ATP) Cohort, which included all evaluable subjects for whom at least one laboratory result of blood sample was available at the survey visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Number analyzed (Participants) | 6401 | 6411 | 6400 | 2399
Participants
  6M-4Y, Overall: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  6M-4Y, Overall | 720 | 574 | 605 | 345
  5-19Y, Overall: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  5-19Y, Overall | 446 | 469 | 483 | 278
  20+Y, Overall: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  20+Y, Overall | 147 | 146 | 193 | 92

2. Secondary Outcome: Number of Subjects With Plasmodium Falciparum (P. Falciparum) Parasitaemia (PFP), According to Annual Age for Children of 4 Years or Less, for Each Survey
Description: The overall parasite prevalence (PP) data were collected across centers from subjects aged 4 years or less, for each Survey. The number of subjects P. Falciparum parasitemia infected among the number of subjects with known result for P.falciparum parasitemia test was tabulated.
Time Frame: At each Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
Participants
  Children aged 0 year: number analyzed (Participants) | 252 | 413 | 334 | 141
  Children aged 0 year | 21 | 38 | 41 | 25
  Children aged 1 year: number analyzed (Participants) | 666 | 722 | 875 | 262
  Children aged 1 year | 94 | 75 | 128 | 62
  Children aged 2 years: number analyzed (Participants) | 628 | 699 | 741 | 305
  Children aged 2 years | 139 | 122 | 125 | 86
  Children aged 3 years: number analyzed (Participants) | 839 | 697 | 635 | 250
  Children aged 3 years | 223 | 174 | 135 | 86
  Children aged 4 years: number analyzed (Participants) | 815 | 666 | 608 | 235
  Children aged 4 years | 243 | 165 | 176 | 86

3. Secondary Outcome: Number of Subjects With Anemia and Severe Anemia for Each Survey
Description: The overall anemia and severe anemia data were collected across centers from subjects, aged between and including: 6M-4Y, 5-19 Y and 20Y+, for each survey. Hemoglobin (Hgb) cut-offs used to define anemia and severe anemia in people living at sea level are: Anemia: children 6M to 5Y, Hgb lower than (<) 11 gram per deciliter (g/dL); children 5-11Y, Hgb <11.5 g/dL; children 12-13Y, Hgb <12 g/dL; non-pregnant females, Hgb <12 g/dL; pregnant females, Hgb <11 g/dL; males, Hgb <13 g/dL. Severe anemia: any age or gender, Hgb <7 g/dL. Missing/ Not applicable (NA) = if age or pregnancy status was not available. Among each age category, results for both sub-categories "Yes" (subjects with anemia) and "Missing/NA" are presented below, results for the category "No" can be deduced from the number of participants analyzed in the corresponding age category, minus (number of "Yes" + number of "Missing/NA"). Similar presentation is followed for "severe anemia" results.
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Number analyzed (Participants) | 6401 | 6411 | 6400 | 2399
Participants
  Overall Yes, Anaemia, 6M-4Y: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  Overall Yes, Anaemia, 6M-4Y | 1974 | 2025 | 1974 | 871
  Missing/NA Anemia, 6M-4Y: number analyzed (Participants) | 3200 | 3197 | 0 | 0
  Missing/NA Anemia, 6M-4Y | 4 | 2 |  |
  Overall Yes, Anemia, 5-19Y: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  Overall Yes, Anemia, 5-19Y | 806 | 794 | 765 | 371
  Missing/NA Anemia, 5-19Y: number analyzed (Participants) | 1613 | 1627 | 0 | 0
  Missing/NA Anemia, 5-19Y | 2 | 2 |  |
  Overall Yes, Anemia, 20Y+: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  Overall Yes, Anemia, 20Y+ | 673 | 631 | 651 | 313
  Missing/NA Anemia, 20Y+: number analyzed (Participants) | 1588 | 1587 | 0 | 0
  Missing/NA Anemia, 20Y+ | 1 | 0 |  |
  Overall Yes, Severe anaemia, 6M-4Y: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  Overall Yes, Severe anaemia, 6M-4Y | 85 | 70 | 84 | 34
  Missing/NA Severe anemia, 6M-4Y: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  Missing/NA Severe anemia, 6M-4Y | 1226 | 1172 | 1219 | 322
  Overall Yes, Severe anaemia, 5-19Y: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  Overall Yes, Severe anaemia, 5-19Y | 10 | 12 | 19 | 5
  Missing/NA Severe anemia, 5-19Y: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  Missing/NA Severe anemia, 5-19Y | 807 | 833 | 847 | 235
  Overall Yes, Severe anaemia, 20Y+: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  Overall Yes, Severe anaemia, 20Y+ | 17 | 14 | 9 | 4
  Missing/NA Severe anemia, 20Y+: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  Missing/NA Severe anemia, 20Y+ | 915 | 956 | 944 | 287

4. Secondary Outcome: Number of Subjects With Anti-malarial Therapy in Survey 1, According to Parasite Density
Description: The overall anti-malaria therapy data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg). Results include the following categories: Malaria treatment (MT) in past 14 days with sub-categories assessed: Yes, No; Exact days of malaria treatment (EDMT) with sub-categories assessed: Ongoing, 1-3 Days, ≥ 4 Days, Missing/NA; Other medication (OM) in past 14 days with sub-categories assessed: Yes, No; Days of other medication (DOM) with sub-categories assessed: Ongoing, 1-7 Days, ≥ 8 Days, Missing/NA; Malaria hospitalization (MH) in the last 3 months with sub-categories assessed: Yes, No. Missing/NA = Missing or Not Applicable.* In case of several medication (malaria treatment or other medication) taken per subject, the maximum duration was computed for this study.
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Low PD Group (Survey 1): Subjects from Survey 1 with low P. falciparum parasite density (PD), (less than [<] 2500 parasites per microliter [parasites/μL]. Infection determined using a blood smear slide and determined using microscopy.
- Medium PD Group (Survey 1): Subjects from Survey 1 with medium P. falciparum parasite density (PD), (2500 - 9999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- High PD Group (Survey 1): Subjects from Survey 1 with high P. falciparum parasite density (PD), (10000 - 19999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Very High PD Group (Survey 1): Subjects from Survey 1 with very high P. falciparum parasite density (PD), (greater than or equal to [≥] 20000 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Neg PD Group (Survey 1): Subjects from Survey 1 not infected with P.falciparum.
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, MT in past 14 days, Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MT in past 14 days, Yes | 22 | 9 | 2 | 12 | 262
  6M-4Y, MT in past 14 days, No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MT in past 14 days, No | 351 | 161 | 56 | 107 | 2218
  6M-4Y, EDMT *, Ongoing: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, EDMT *, Ongoing | 3 | 2 | 0 | 0 | 28
  6M-4Y, EDMT *, 1-3 days: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, EDMT *, 1-3 days | 18 | 5 | 2 | 9 | 206
  6M-4Y, EDMT *, ≥ 4days: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, EDMT *, ≥ 4days | 1 | 2 | 0 | 3 | 27
  6M-4Y, EDMT *, Missing/Not applicable: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, EDMT *, Missing/Not applicable | 351 | 161 | 56 | 107 | 2219
  6M-4Y, OM in past 14 days, Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, OM in past 14 days, Yes | 35 | 33 | 21 | 33 | 445
  6M-4Y, OM in past 14 days, No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, OM in past 14 days, No | 338 | 137 | 37 | 86 | 2035
  6M-4Y, DOM *, Ongoing: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, DOM *, Ongoing | 8 | 7 | 2 | 5 | 79
  6M-4Y, DOM *, 1-7 days: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, DOM *, 1-7 days | 25 | 26 | 19 | 27 | 365
  6M-4Y, DOM *, ≥ 8 days: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 1
  6M-4Y, DOM *, Missing/Not applicable: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, DOM *, Missing/Not applicable | 340 | 137 | 37 | 87 | 2035
  6M-4Y, MH in the last 3 months, Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MH in the last 3 months, Yes | 7 | 4 | 1 | 7 | 90
  6M-4Y, MH in the last 3 months, No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MH in the last 3 months, No | 366 | 166 | 57 | 112 | 2390
  5-19Y, MT in past 14 days, Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MT in past 14 days, Yes | 5 | 6 | 4 | 2 | 85
  5-19Y, MT in past 14 days, No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MT in past 14 days, No | 289 | 65 | 19 | 56 | 1082
  5-19Y, EDMT *, Ongoing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, EDMT *, Ongoing | 1 | 0 | 0 | 0 | 5
  5-19Y, EDMT *, 1-3 days: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, EDMT *, 1-3 days | 4 | 6 | 4 | 1 | 75
  5-19Y, EDMT *, ≥ 4days: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, EDMT *, ≥ 4days | 0 | 0 | 0 | 1 | 5
  5-19Y, EDMT *, Missing/Not applicable: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, EDMT *, Missing/Not applicable | 289 | 65 | 19 | 56 | 1082
  5-19Y, OM in past 14 days, Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, OM in past 14 days, Yes | 29 | 12 | 8 | 7 | 143
  5-19Y, OM in past 14 days, No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, OM in past 14 days, No | 265 | 59 | 15 | 51 | 1024
  5-19Y, DOM *, Ongoing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, DOM *, Ongoing | 4 | 1 | 1 | 2 | 17
  5-19Y, DOM *, 1-7 days: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, DOM *, 1-7 days | 25 | 11 | 7 | 5 | 125
  5-19Y, DOM *, ≥ 8 days: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 0
  5-19Y, DOM *, Missing/Not applicable: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, DOM *, Missing/Not applicable | 265 | 59 | 15 | 51 | 1025
  5-19Y, MH in the last 3 months, Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MH in the last 3 months, Yes | 0 | 3 | 0 | 1 | 24
  5-19Y, MH in the last 3 months, No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MH in the last 3 months, No | 294 | 68 | 23 | 57 | 1143
  20Y+, MT in past 14 days, Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, MT in past 14 days, Yes | 1 | 0 |  | 0 | 102
  20Y+, MT in past 14 days, No: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, MT in past 14 days, No | 118 | 17 |  | 11 | 1339
  20Y+, EDMT *, Ongoing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, EDMT *, Ongoing | 0 | 0 |  | 0 | 14
  20Y+, EDMT *, 1-3 days: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, EDMT *, 1-3 days | 1 | 0 |  | 0 | 80
  20Y+, EDMT *, ≥ 4days: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, EDMT *, ≥ 4days | 0 | 0 |  | 0 | 8
  20Y+, EDMT *, Missing/Not applicable: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, EDMT *, Missing/Not applicable | 118 | 17 |  | 11 | 1339
  20Y+, OM in past 14 days, Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, OM in past 14 days, Yes | 20 | 6 |  | 2 | 203
  20Y+, OM in past 14 days, No: number analyzed (Participants) | 119 | 17 | 0 | 188 | 1441
  20Y+, OM in past 14 days, No | 99 | 11 |  | 9 | 1238
  20Y+, DOM *, Ongoing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, DOM *, Ongoing | 5 | 1 |  | 1 | 41
  20Y+, DOM *, 1-7 days: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, DOM *, 1-7 days | 15 | 5 |  | 1 | 158
  20Y+, DOM *, ≥ 8 days: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, DOM *, ≥ 8 days | 0 | 0 |  | 0 | 2
  20Y+, DOM *, Missing/Not applicable: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, DOM *, Missing/Not applicable | 99 | 11 |  | 9 | 1240
  20Y+, MH in the last 3 months, Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, MH in the last 3 months, Yes | 0 | 2 |  | 0 | 18
  20Y+, MH in the last 3 months, No: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20Y+, MH in the last 3 months, No | 119 | 15 |  | 11 | 1423

5. Secondary Outcome: Number of Subjects With Anti-malarial Therapy in Survey 2, According to Parasite Density
Description: The overall anti-malaria therapy data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg). Results include the following categories: Malaria treatment (MT) in past 14 days with sub-categories assessed: Yes, No; Exact days of malaria treatment (EDMT) with sub-categories assessed: Ongoing, 1-3 Days, ≥ 4 Days, Missing/NA; Other medication (OM) in past 14 days with sub-categories assessed: Yes, No; Days of other medication (DOM) with sub-categories assessed: Ongoing, 1-7 Days, ≥ 8 Days, Missing/NA; Malaria hospitalization (MH) in the last 3 months with sub-categories assessed: Yes, No. Missing/NA = Missing or Not Applicable.* In case of several medication (malaria treatment or other medication) taken per subject, the maximum duration was computed for this study.
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Low PD Group (Survey 2): Subjects from Survey 2 with low P. falciparum parasite density (PD), (less than [<] 2500 parasites per microliter [parasites/μL]. Infection determined using a blood smear slide and determined using microscopy.
- Medium PD Group (Survey 2): Subjects from Survey 2 with medium P. falciparum parasite density (PD), (2500 - 9999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- High PD Group (Survey 2): Subjects from Survey 2 with high P. falciparum parasite density (PD), (10000 - 19999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Very High PD Group (Survey 2): Subjects from Survey 2 with very high P. falciparum parasite density (PD), (greater than or equal to [≥] 20000 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Neg PD Group (Survey 2): Subjects from Survey 2 not infected with P.falciparum.
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, MT in past 14 days, Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MT in past 14 days, Yes | 14 | 6 | 2 | 5 | 257
  6M-4Y, MT in past 14 days, No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MT in past 14 days, No | 269 | 142 | 65 | 71 | 2366
  6M-4Y, EDMT *, Ongoing: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, EDMT *, Ongoing | 1 | 3 | 0 | 1 | 25
  6M-4Y, EDMT *, 1-3 days: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, EDMT *, 1-3 days | 12 | 1 | 1 | 4 | 206
  6M-4Y, EDMT *, ≥ 4days: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, EDMT *, ≥ 4days | 1 | 2 | 1 | 0 | 26
  6M-4Y, EDMT *, Missing/NA: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, EDMT *, Missing/NA | 269 | 142 | 65 | 71 | 2366
  6M-4Y, OM in past 14 days, Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, OM in past 14 days, Yes | 42 | 15 | 9 | 17 | 535
  6M-4Y, OM in past 14 days, No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, OM in past 14 days, No | 241 | 133 | 58 | 59 | 2088
  6M-4Y, DOM *, Ongoing: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, DOM *, Ongoing | 12 | 6 | 3 | 2 | 118
  6M-4Y, DOM *, 1-7 days: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, DOM *, 1-7 days | 30 | 9 | 6 | 15 | 410
  6M-4Y, DOM *, ≥ 8 days: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 7
  6M-4Y, DOM *, Missing/NA: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, DOM *, Missing/NA | 241 | 133 | 58 | 59 | 2088
  6M-4Y, MH in the last 3 months, Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MH in the last 3 months, Yes | 3 | 3 | 2 | 3 | 77
  6M-4Y, MH in the last 3 months, No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MH in the last 3 months, No | 280 | 145 | 65 | 73 | 2546
  5-19Y, MT in past 14 days, Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MT in past 14 days, Yes | 11 | 3 | 2 | 4 | 77
  5-19Y, MT in past 14 days, No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MT in past 14 days, No | 322 | 68 | 27 | 32 | 1081
  5-19Y, EDMT *, Ongoing: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, EDMT *, Ongoing | 1 | 1 | 0 | 0 | 11
  5-19Y, EDMT *, 1-3 days: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, EDMT *, 1-3 days | 8 | 1 | 2 | 4 | 66
  5-19Y, EDMT *, ≥ 4days: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, EDMT *, ≥ 4days | 2 | 1 | 0 | 0 | 0
  5-19Y, EDMT *, Missing/NA: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, EDMT *, Missing/NA | 322 | 68 | 27 | 32 | 1081
  5-19Y, OM in past 14 days, Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, OM in past 14 days, Yes | 33 | 10 | 8 | 9 | 134
  5-19Y, OM in past 14 days, No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, OM in past 14 days, No | 300 | 61 | 21 | 27 | 1024
  5-19Y, DOM *, Ongoing: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, DOM *, Ongoing | 7 | 1 | 0 | 1 | 30
  5-19Y, DOM *, 1-7 days: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, DOM *, 1-7 days | 26 | 9 | 8 | 8 | 102
  5-19Y, DOM *, ≥ 8 days: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 2
  5-19Y, DOM *, Missing/NA: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, DOM *, Missing/NA | 300 | 61 | 21 | 27 | 1024
  5-19Y, MH in the last 3 months, Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MH in the last 3 months, Yes | 5 | 1 | 1 | 1 | 19
  5-19Y, MH in the last 3 months, No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MH in the last 3 months, No | 328 | 70 | 28 | 35 | 1139
  20Y+, MT in past 14 days, Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, MT in past 14 days, Yes | 2 | 0 | 0 | 2 | 84
  20Y+, MT in past 14 days, No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, MT in past 14 days, No | 122 | 10 | 5 | 5 | 1357
  20Y+, EDMT *, Ongoing: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, EDMT *, Ongoing | 0 | 0 | 0 | 1 | 5
  20Y+, EDMT *, 1-3 days: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, EDMT *, 1-3 days | 2 | 0 | 0 | 1 | 72
  20Y+, EDMT *, ≥ 4days: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, EDMT *, ≥ 4days | 0 | 0 | 0 | 0 | 7
  20Y+, EDMT *, Missing/NA: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, EDMT *, Missing/NA | 122 | 10 | 5 | 5 | 1357
  20Y+, OM in past 14 days, Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, OM in past 14 days, Yes | 10 | 2 | 2 | 3 | 214
  20Y+, OM in past 14 days, No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, OM in past 14 days, No | 114 | 8 | 3 | 4 | 1227
  20Y+, DOM *, Ongoing: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, DOM *, Ongoing | 1 | 0 | 1 | 2 | 71
  20Y+, DOM *, 1-7 days: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, DOM *, 1-7 days | 9 | 2 | 1 | 1 | 138
  20Y+, DOM *, ≥ 8 days: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 5
  20Y+, DOM *, Missing/NA: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, DOM *, Missing/NA | 114 | 8 | 3 | 4 | 1227
  20Y+, MH in the last 3 months, Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, MH in the last 3 months, Yes | 1 | 1 | 0 | 0 | 19
  20Y+, MH in the last 3 months, No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20Y+, MH in the last 3 months, No | 123 | 9 | 5 | 7 | 1422

6. Secondary Outcome: Number of Subjects With Anti-malarial Therapy in Survey 3, According to Parasite Density
Description: The overall anti-malaria therapy data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg). Results include the following categories: Malaria treatment (MT) in past 14 days with sub-categories assessed: Yes, No; Exact days of malaria treatment (EDMT) with sub-categories assessed: Ongoing, 1-3 Days, ≥ 4 Days, Missing/NA; Other medication (OM) in past 14 days with sub-categories assessed: Yes, No; Days of other medication (DOM) with sub-categories assessed: Ongoing, 1-7 Days, ≥ 8 Days, Missing/NA; Malaria hospitalization (MH) in the last 3 months with sub-categories assessed: Yes, No. Missing/NA = Missing or Not Applicable.* In case of several medication (malaria treatment or other medication) taken per subject, the maximum duration was computed for this study.
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Low PD Group (Survey 3): Subjects from Survey 3 with low P. falciparum parasite density (PD), (less than [<] 2500 parasites per microliter [parasites/μL]. Infection determined using a blood smear slide and determined using microscopy.
- Medium PD Group (Survey 3): Subjects from Survey 3 with medium P. falciparum parasite density (PD), (2500 - 9999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- High PD Group (Survey 3): Subjects from Survey 3 with high P. falciparum parasite density (PD), (10000 - 19999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Very High PD Group (Survey 3): Subjects from Survey 3 with very high P. falciparum parasite density (PD), (greater than or equal to [≥] 20000 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Neg PD Group (Survey 3): Subjects from Survey 3 not infected with P.falciparum.
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, MT in past 14 days, Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MT in past 14 days, Yes | 17 | 13 | 3 | 9 | 267
  6M-4Y, MT in past 14 days, No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MT in past 14 days, No | 262 | 148 | 71 | 82 | 2321
  6M-4Y, EDMT *, Ongoing: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, EDMT *, Ongoing | 4 | 1 | 0 | 4 | 33
  6M-4Y, EDMT *, 1-3 days: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, EDMT *, 1-3 days | 11 | 10 | 3 | 5 | 210
  6M-4Y, EDMT *, ≥ 4days: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, EDMT *, ≥ 4days | 2 | 2 | 0 | 0 | 24
  6M-4Y, EDMT *, Missing/NA: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, EDMT *, Missing/NA | 262 | 148 | 71 | 82 | 2321
  6M-4Y, OM in past 14 days, Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, OM in past 14 days, Yes | 65 | 30 | 18 | 18 | 547
  6M-4Y, OM in past 14 days, No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, OM in past 14 days, No | 214 | 131 | 56 | 73 | 2041
  6M-4Y, DOM *, Ongoing: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, DOM *, Ongoing | 10 | 8 | 3 | 6 | 142
  6M-4Y, DOM *, 1-7 days: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, DOM *, 1-7 days | 55 | 22 | 15 | 12 | 394
  6M-4Y, DOM *, ≥ 8 days: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 11
  6M-4Y, DOM *, Missing/NA: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, DOM *, Missing/NA | 214 | 131 | 56 | 73 | 2041
  6M-4Y, MH in the last 3 months, Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MH in the last 3 months, Yes | 14 | 4 | 3 | 0 | 99
  6M-4Y, MH in the last 3 months, No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MH in the last 3 months, No | 265 | 157 | 71 | 91 | 2489
  5-19Y, MT in past 14 days, Yes: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MT in past 14 days, Yes | 14 | 4 | 1 | 1 | 58
  5-19Y, MT in past 14 days, No: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MT in past 14 days, No | 327 | 90 | 12 | 34 | 1071
  5-19Y, EDMT *, Ongoing: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, EDMT *, Ongoing | 4 | 1 | 0 | 0 | 4
  5-19Y, EDMT *, 1-3 days: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, EDMT *, 1-3 days | 8 | 3 | 1 | 1 | 50
  5-19Y, EDMT *, ≥ 4days: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, EDMT *, ≥ 4days | 2 | 0 | 0 | 0 | 4
  5-19Y, EDMT *, Missing/NA: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, EDMT *, Missing/NA | 327 | 90 | 12 | 34 | 1071
  5-19Y, OM in past 14 days, Yes: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, OM in past 14 days, Yes | 44 | 18 | 3 | 13 | 128
  5-19Y, OM in past 14 days, No: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, OM in past 14 days, No | 297 | 76 | 10 | 22 | 1001
  5-19Y, DOM *, Ongoing: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, DOM *, Ongoing | 13 | 1 | 0 | 2 | 19
  5-19Y, DOM *, 1-7 days: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, DOM *, 1-7 days | 31 | 17 | 3 | 11 | 109
  5-19Y, DOM *, ≥ 8 days: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 0
  5-19Y, DOM *, Missing/NA: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, DOM *, Missing/NA | 297 | 76 | 10 | 22 | 1001
  5-19Y, MH in the last 3 months, Yes: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MH in the last 3 months, Yes | 7 | 0 | 0 | 1 | 17
  5-19Y, MH in the last 3 months, No: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MH in the last 3 months, No | 334 | 94 | 13 | 34 | 1112
  20Y+, MT in past 14 days, Yes: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, MT in past 14 days, Yes | 5 | 2 | 0 | 0 | 70
  20Y+, MT in past 14 days, No: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, MT in past 14 days, No | 166 | 11 | 5 | 4 | 1332
  20Y+, EDMT *, Ongoing: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, EDMT *, Ongoing | 0 | 0 | 0 | 0 | 6
  20Y+, EDMT *, 1-3 days: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, EDMT *, 1-3 days | 5 | 1 | 0 | 0 | 63
  20Y+, EDMT *, ≥ 4days: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, EDMT *, ≥ 4days | 0 | 1 | 0 | 0 | 1
  20Y+, EDMT *, Missing/NA: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, EDMT *, Missing/NA | 166 | 11 | 5 | 4 | 1332
  20Y+, OM in past 14 days, Yes: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, OM in past 14 days, Yes | 25 | 3 | 3 | 1 | 227
  20Y+, OM in past 14 days, No: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, OM in past 14 days, No | 146 | 10 | 2 | 3 | 1175
  20Y+, DOM *, Ongoing: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, DOM *, Ongoing | 5 | 3 | 0 | 1 | 70
  20Y+, DOM *, 1-7 days: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, DOM *, 1-7 days | 19 | 0 | 3 | 0 | 151
  20Y+, DOM *, ≥ 8 days: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, DOM *, ≥ 8 days | 1 | 0 | 0 | 0 | 6
  20Y+, DOM *, Missing/NA: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, DOM *, Missing/NA | 146 | 10 | 2 | 3 | 1175
  20Y+, MH in the last 3 months, Yes: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, MH in the last 3 months, Yes | 0 | 0 | 0 | 0 | 12
  20Y+, MH in the last 3 months, No: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20Y+, MH in the last 3 months, No | 171 | 13 | 5 | 4 | 1390

7. Secondary Outcome: Number of Subjects With Anti-malarial Therapy in Survey 4, According to Parasite Density
Description: The overall anti-malaria therapy data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg). Results include the following categories: Malaria treatment (MT) in past 14 days with sub-categories assessed: Yes, No; Exact days of malaria treatment (EDMT) with sub-categories assessed: Ongoing, 1-3 Days, ≥ 4 Days, Missing/NA; Other medication (OM) in past 14 days with sub-categories assessed: Yes, No; Days of other medication (DOM) with sub-categories assessed: Ongoing, 1-7 Days, ≥ 8 Days, Missing/NA; Malaria hospitalization (MH) in the last 3 months with sub-categories assessed: Yes, No. Missing/NA = Missing or Not Applicable.* In case of several medication (malaria treatment or other medication) taken per subject, the maximum duration was computed for this study.
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Low PD Group (Survey 4): Subjects from Survey 4 with low P. falciparum parasite density (PD), (less than [<] 2500 parasites per microliter [parasites/μL]. Infection determined using a blood smear slide and determined using microscopy.
- Medium PD Group (Survey 4): Subjects from Survey 4 with medium P. falciparum parasite density (PD), (2500 - 9999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- High PD Group (Survey 4): Subjects from Survey 4 with high P. falciparum parasite density (PD), (10000 - 19999 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Very High PD Group (Survey 4): Subjects from Survey 4 with very high P. falciparum parasite density (PD), (greater than or equal to [≥] 20000 parasites/μL). Infection determined using a blood smear slide and determined using microscopy.
- Neg PD Group (Survey 4): Subjects from Survey 4 not infected with P.falciparum.
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, MT in past 14 days, Yes: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, MT in past 14 days, Yes | 5 | 2 | 1 | 5 | 71
  6M-4Y, MT in past 14 days, No: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, MT in past 14 days, No | 163 | 101 | 19 | 49 | 777
  6M-4Y, EDMT *, Ongoing: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, EDMT *, Ongoing | 2 | 1 | 0 | 4 | 21
  6M-4Y, EDMT *, 1-3 days: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, EDMT *, 1-3 days | 3 | 1 | 1 | 1 | 49
  6M-4Y, EDMT *, ≥ 4days: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, EDMT *, ≥ 4days | 0 | 0 | 0 | 0 | 1
  6M-4Y, EDMT *, Missing/NA: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, EDMT *, Missing/NA | 163 | 101 | 19 | 49 | 777
  6M-4Y, OM in past 14 days, Yes: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, OM in past 14 days, Yes | 21 | 11 | 7 | 12 | 152
  6M-4Y, OM in past 14 days, No: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, OM in past 14 days, No | 147 | 92 | 13 | 42 | 696
  6M-4Y, DOM *, Ongoing: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, DOM *, Ongoing | 5 | 2 | 3 | 5 | 48
  6M-4Y, DOM *, 1-7 days: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, DOM *, 1-7 days | 16 | 8 | 4 | 7 | 103
  6M-4Y, DOM *, ≥ 8 days: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, DOM *, ≥ 8 days | 0 | 1 | 0 | 0 | 1
  6M-4Y, DOM *, Missing/NA: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, DOM *, Missing/NA | 147 | 92 | 13 | 42 | 696
  6M-4Y, MH in the last 3 months, Yes: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, MH in the last 3 months, Yes | 9 | 1 | 0 | 2 | 28
  6M-4Y, MH in the last 3 months, No: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, MH in the last 3 months, No | 159 | 102 | 20 | 52 | 820
  5-19Y, MT in past 14 days, Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MT in past 14 days, Yes | 2 | 0 | 0 | 0 | 10
  5-19Y, MT in past 14 days, No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MT in past 14 days, No | 196 | 51 | 16 | 13 | 318
  5-19Y, EDMT *, Ongoing: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, EDMT *, Ongoing | 0 | 0 | 0 | 0 | 3
  5-19Y, EDMT *, 1-3 days: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, EDMT *, 1-3 days | 2 | 0 | 0 | 0 | 7
  5-19Y, EDMT *, ≥ 4days: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, EDMT *, ≥ 4days | 0 | 0 | 0 | 0 | 0
  5-19Y, EDMT *, Missing/NA: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, EDMT *, Missing/NA | 196 | 51 | 16 | 13 | 318
  5-19Y, OM in past 14 days, Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, OM in past 14 days, Yes | 13 | 4 | 0 | 2 | 28
  5-19Y, OM in past 14 days, No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, OM in past 14 days, No | 185 | 47 | 16 | 11 | 300
  5-19Y, DOM *, Ongoing: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, DOM *, Ongoing | 1 | 0 | 0 | 1 | 6
  5-19Y, DOM *, 1-7 days: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, DOM *, 1-7 days | 12 | 4 | 0 | 1 | 22
  5-19Y, DOM *, ≥ 8 days: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, DOM *, ≥ 8 days | 0 | 0 | 0 | 0 | 0
  5-19Y, DOM *, Missing/NA: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, DOM *, Missing/NA | 185 | 47 | 16 | 11 | 300
  5-19Y, MH in the last 3 months, Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MH in the last 3 months, Yes | 0 | 0 | 0 | 0 | 2
  5-19Y, MH in the last 3 months, No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MH in the last 3 months, No | 198 | 51 | 16 | 13 | 326
  20Y+, MT in past 14 days, Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, MT in past 14 days, Yes | 1 | 0 |  | 0 | 8
  20Y+, MT in past 14 days, No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, MT in past 14 days, No | 86 | 4 |  | 1 | 500
  20Y+, EDMT *, Ongoing: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, EDMT *, Ongoing | 0 | 0 |  | 0 | 1
  20Y+, EDMT *, 1-3 days: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, EDMT *, 1-3 days | 1 | 0 |  | 0 | 5
  20Y+, EDMT *, ≥ 4days: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, EDMT *, ≥ 4days | 0 | 0 |  | 0 | 2
  20Y+, EDMT *, Missing/NA: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, EDMT *, Missing/NA | 86 | 4 |  | 1 | 500
  20Y+, OM in past 14 days, Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, OM in past 14 days, Yes | 5 | 0 |  | 0 | 57
  20Y+, OM in past 14 days, No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, OM in past 14 days, No | 82 | 4 |  | 1 | 451
  20Y+, DOM *, Ongoing: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, DOM *, Ongoing | 1 | 0 |  | 0 | 18
  20Y+, DOM *, 1-7 days: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, DOM *, 1-7 days | 4 | 0 |  | 0 | 36
  20Y+, DOM *, ≥ 8 days: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, DOM *, ≥ 8 days | 0 | 0 |  | 0 | 3
  20Y+, DOM *, Missing/NA: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, DOM *, Missing/NA | 82 | 4 |  | 1 | 451
  20Y+, MH in the last 3 months, Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, MH in the last 3 months, Yes | 0 | 0 |  | 0 | 5
  20Y+, MH in the last 3 months, No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20Y+, MH in the last 3 months, No | 87 | 4 |  | 1 | 503

8. Secondary Outcome: Mean Number of Days With Malaria Treatment at Survey 1
Description: The mean and standard deviation of the number of days of malaria treatment (DMT) were calculated for the past 14 days period of treatment. The malaria treatment data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the 14 day-period before the malaria treatment
Population: Analysis was performed on the According-to-Protocol (ATP) Cohort, which included all evaluable subjects for whom at least one laboratory result of blood sample was available at the survey visit and who have data available during the past 14 days period of Malaria treatment.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 24 | 13 | 6 | 14 | 401
Days
  6M-4Y, DMT: number analyzed (Participants) | 19 | 7 | 2 | 12 | 233
  6M-4Y, DMT | 2.6 (1.02) | 3.7 (1.70) | 2.5 (0.71) | 3.1 (0.67) | 3.1 (1.45)
  5-19Y, DMT: number analyzed (Participants) | 4 | 6 | 4 | 2 | 80
  5-19Y, DMT | 2.0 (0.82) | 2.2 (0.98) | 2.8 (0.50) | 3.5 (0.71) | 2.5 (1.09)
  20+Y, DMT: number analyzed (Participants) | 1 | 0 | 0 | 0 | 88
  20+Y, DMT | 1.0 (0.00) |  |  |  | 2.6 (1.37)

9. Secondary Outcome: Mean Number of Days With Malaria Treatment at Survey 2
Description: The mean and standard deviation of the number of days of malaria treatment (DMT) were calculated for the past 14 days period of treatment. The malaria treatment data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the 14 day-period before the malaria treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 25 | 5 | 4 | 9 | 377
Days
  6M-4Y, DMT: number analyzed (Participants) | 13 | 3 | 2 | 4 | 232
  6M-4Y, DMT | 2.8 (1.48) | 5.7 (2.31) | 3.5 (0.71) | 2.0 (1.15) | 3.1 (1.16)
  5-19Y, DMT: number analyzed (Participants) | 10 | 2 | 2 | 4 | 66
  5-19Y, DMT | 2.8 (1.81) | 3.5 (2.12) | 3.0 (0.00) | 2.5 (1.00) | 2.5 (0.81)
  20+Y, DMT: number analyzed (Participants) | 2 | 0 | 0 | 1 | 79
  20+Y, DMT | 3.0 (0.00) |  |  | 1.0 (0.00) | 2.5 (1.37)

10. Secondary Outcome: Mean Number of Days With Malaria Treatment at Survey 3
Description: The mean and standard deviation of the number of days of malaria treatment (DMT) were calculated for the past 14 days period of treatment. The malaria treatment data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the 14 day-period before the malaria treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 28 | 17 | 4 | 6 | 352
Days
  6M-4Y, DMT: number analyzed (Participants) | 13 | 12 | 3 | 5 | 234
  6M-4Y, DMT | 3.0 (0.71) | 3.3 (1.07) | 2.3 (1.15) | 2.2 (1.10) | 3.1 (1.08)
  5-19Y, DMT: number analyzed (Participants) | 10 | 3 | 1 | 1 | 54
  5-19Y, DMT | 3.9 (2.88) | 1.7 (1.15) | 3.0 (0.00) | 1.0 (0.00) | 2.9 (1.27)
  20+Y, DMT: number analyzed (Participants) | 5 | 2 | 0 | 0 | 64
  20+Y, DMT | 1.4 (0.89) | 5.0 (2.83) |  |  | 2.3 (1.12)

11. Secondary Outcome: Mean Number of Days With Malaria Treatment at Survey 4
Description: The mean and standard deviation of the number of days of malaria treatment (DMT) were calculated for the past 14 days period of treatment. The malaria treatment data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the 14 day-period before the malaria treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 6 | 1 | 1 | 1 | 64
Days
  6M-4Y, DMT: number analyzed (Participants) | 3 | 1 | 1 | 1 | 50
  6M-4Y, DMT | 2.3 (1.15) | 3.0 (0.00) | 3.0 (0.00) | 1.0 (0.00) | 3.1 (0.59)
  5-19Y, DMT: number analyzed (Participants) | 2 | 0 | 0 | 0 | 7
  5-19Y, DMT | 3.0 (0.00) |  |  |  | 2.9 (0.38)
  20+Y, DMT: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7
  20+Y, DMT | 1.0 (0.00) |  |  |  | 3.3 (2.14)

12. Secondary Outcome: Number of Subjects With Fever in the Last 24 Hours or at Visit During Survey 1
Description: Measured characteristics of fever were the following: Fever in the last 24 hours (F 24h) and Fever at visit (F at V). Note: Fever set to "Yes" if temperature recorded after axillary conversion was ≥ 37.5 degrees Celsius (°C). Missing/NA = Missing or Not Applicable. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: In the last 24 hours or at the survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, F 24h - Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, F 24h - Yes | 71 | 53 | 21 | 60 | 361
  6M-4Y, F 24h - No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, F 24h - No | 302 | 117 | 37 | 59 | 2119
  6M-4Y, F at V - Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, F at V - Yes | 26 | 13 | 7 | 22 | 79
  6M-4Y, F at V - No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, F at V - No | 347 | 157 | 51 | 97 | 2400
  6M-4Y, F at V - Missing/NA: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, F at V - Missing/NA | 0 | 0 | 0 | 0 | 1
  5-19Y, F 24h - Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, F 24h - Yes | 37 | 25 | 10 | 24 | 124
  5-19Y, F 24h - No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, F 24h - No | 257 | 46 | 13 | 34 | 1043
  5-19Y, F at V - Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, F at V - Yes | 6 | 5 | 5 | 17 | 29
  5-19Y, F at V - No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, F at V - No | 288 | 66 | 18 | 41 | 1138
  20+Y, F 24h - Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, F 24h - Yes | 30 | 9 |  | 2 | 181
  20+Y, F 24h - No: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, F 24h - No | 89 | 8 |  | 9 | 1260
  20+Y, F at V - Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, F at V - Yes | 3 | 0 |  | 1 | 23
  20+Y, F at V - No: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, F at V - No | 115 | 17 |  | 10 | 1418
  20+Y, F at V - Missing/NA: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, F at V - Missing/NA | 1 | 0 |  | 0 | 0

13. Secondary Outcome: Number of Subjects With Fever in the Last 24 Hours or at Visit During Survey 2
Description: Measured characteristics of fever were the following: Fever in the last 24 hours (F 24h) and Fever at visit (F at V). Note: Fever set to "Yes" if temperature recorded after axillary conversion was ≥ 37.5 degrees Celsius (°C). Missing/NA = Missing or Not Applicable. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: In the last 24 hours or at the survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, F 24h - Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, F 24h - Yes | 41 | 23 | 15 | 35 | 357
  6M-4Y, F 24h - No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, F 24h - No | 242 | 125 | 52 | 41 | 2266
  6M-4Y, F at V - Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, F at V - Yes | 26 | 16 | 15 | 29 | 98
  6M-4Y, F at V - No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, F at V - No | 257 | 132 | 52 | 47 | 2525
  5-19Y, F 24h - Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, F 24h - Yes | 39 | 11 | 11 | 13 | 115
  5-19Y, F 24h - No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, F 24h - No | 294 | 60 | 18 | 23 | 1043
  5-19Y, F at V - Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, F at V - Yes | 24 | 4 | 3 | 8 | 26
  5-19Y, F at V - No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, F at V - No | 309 | 67 | 26 | 28 | 1132
  20+Y, F 24h - Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, F 24h - Yes | 14 | 4 | 3 | 2 | 169
  20+Y, F 24h - No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, F 24h - No | 110 | 6 | 2 | 5 | 1272
  20+Y, F at V - Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, F at V - Yes | 10 | 0 | 0 | 1 | 36
  20+Y, F at V - No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, F at V - No | 114 | 10 | 5 | 6 | 1404
  20+Y, F at V - Missing/NA: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, F at V - Missing/NA | 0 | 0 | 0 | 0 | 1

14. Secondary Outcome: Number of Subjects With Fever in the Last 24 Hours or at Visit During Survey 3
Description: Measured characteristics of fever were the following: Fever in the last 24 hours (F 24h) and Fever at visit (F at V). Note: Fever set to "Yes" if temperature recorded after axillary conversion was ≥ 37.5 degrees Celsius (°C). Missing/NA = Missing or Not Applicable. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: In the last 24 hours or at the survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, F 24h - Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, F 24h - Yes | 60 | 44 | 28 | 44 | 360
  6M-4Y, F 24h - No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, F 24h - No | 219 | 117 | 46 | 47 | 2228
  6M-4Y, F at V - Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, F at V - Yes | 8 | 16 | 9 | 22 | 56
  6M-4Y, F at V - No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, F at V - No | 271 | 145 | 65 | 69 | 2532
  5-19Y, F 24h - Yes: number analyzed (Participants) | 341 | 93 | 13 | 35 | 1129
  5-19Y, F 24h - Yes | 54 | 25 | 4 | 17 | 92
  5-19Y, F 24h - No: number analyzed (Participants) | 341 | 93 | 13 | 35 | 1129
  5-19Y, F 24h - No | 287 | 69 | 9 | 18 | 1037
  5-19Y, F at V - Yes: number analyzed (Participants) | 341 | 93 | 13 | 35 | 1129
  5-19Y, F at V - Yes | 11 | 6 | 1 | 14 | 21
  5-19Y, F at V - No: number analyzed (Participants) | 341 | 93 | 13 | 35 | 1129
  5-19Y, F at V - No | 330 | 87 | 12 | 21 | 1107
  5-19Y, F at V - Missing/NA: number analyzed (Participants) | 171 | 14 | 5 | 4 | 1403
  5-19Y, F at V - Missing/NA | 0 | 1 | 0 | 0 | 1
  20+Y, F 24h - Yes: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, F 24h - Yes | 20 | 4 | 4 | 1 | 167
  20+Y, F 24h - No: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, F 24h - No | 151 | 9 | 1 | 3 | 1235
  20+Y, F at V - Yes: number analyzed (Participants) | 171 | 14 | 5 | 4 | 1403
  20+Y, F at V - Yes | 5 | 0 | 3 | 1 | 23
  20+Y, F at V - No: number analyzed (Participants) | 171 | 14 | 5 | 4 | 1403
  20+Y, F at V - No | 166 | 13 | 2 | 3 | 1378
  20+Y, F at V - Missing/NA: number analyzed (Participants) | 171 | 14 | 5 | 4 | 1403
  20+Y, F at V - Missing/NA | 0 | 0 | 0 | 0 | 1

15. Secondary Outcome: Number of Subjects With Fever in the Last 24 Hours or at Visit During Survey 4
Description: Measured characteristics of fever were the following: Fever in the last 24 hours (F 24h) and Fever at visit (F at V). Note: Fever set to "Yes" if temperature recorded after axillary conversion was ≥ 37.5 degrees Celsius (°C). Missing/NA = Missing or Not Applicable. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: In the last 24 hours or at the survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, F 24h - Yes: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, F 24h - Yes | 39 | 18 | 5 | 27 | 115
  6M-4Y, F 24h - No: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, F 24h - No | 129 | 85 | 15 | 27 | 733
  6M-4Y, F at V - Yes: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, F at V - Yes | 8 | 8 | 4 | 18 | 20
  6M-4Y, F at V - No: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, F at V - No | 160 | 95 | 16 | 36 | 827
  6M-4Y, F at V - Missing/NA: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, F at V - Missing/NA | 0 | 0 | 0 | 0 | 1
  5-19Y, F 24h - Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, F 24h - Yes | 38 | 8 | 4 | 4 | 22
  5-19Y, F 24h - No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, F 24h - No | 160 | 43 | 12 | 9 | 306
  5-19Y, F at V - Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, F at V - Yes | 5 | 0 | 2 | 1 | 4
  5-19Y, F at V - No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, F at V - No | 193 | 51 | 14 | 12 | 324
  20+Y, F 24h - Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, F 24h - Yes | 11 | 0 |  | 0 | 25
  20+Y, F 24h - No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, F 24h - No | 76 | 4 |  | 1 | 483
  20+Y, F at V - Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, F at V - Yes | 0 | 0 |  | 0 | 3
  20+Y, F at V - No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, F at V - No | 87 | 4 |  | 1 | 505

16. Secondary Outcome: Mean Number of Days With Fever at Survey 1
Description: The mean and standard deviation of the number of days ago with fever start (DaFs) were calculated for subjects having fever in the last 24 hours. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the survey period (approximatively 1 year)
Population: Analysis was performed on the According-to-Protocol (ATP) Cohort, which included all evaluable subjects for whom at least one laboratory result of blood sample was available at the survey visit and with fever reported in the last 24 hours.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 138 | 87 | 31 | 86 | 663
Days
  6M-4Y, DaFs: number analyzed (Participants) | 71 | 53 | 21 | 60 | 360
  6M-4Y, DaFs | 2.5 (2.18) | 2.6 (2.23) | 2.1 (1.42) | 2.5 (4.13) | 2.3 (1.77)
  5-19Y, DaFs: number analyzed (Participants) | 37 | 25 | 10 | 24 | 124
  5-19Y, DaFs | 2.2 (1.41) | 2.2 (1.29) | 2.7 (2.06) | 1.7 (1.05) | 2.3 (1.93)
  20+Y, DaFs: number analyzed (Participants) | 30 | 9 | 0 | 2 | 179
  20+Y, DaFs | 2.3 (1.56) | 2.3 (1.87) |  | 2.5 (0.71) | 2.9 (3.36)

17. Secondary Outcome: Mean Number of Days With Fever at Survey 2
Description: The mean and standard deviation of the number of days ago with fever start (DaFs) were calculated for subjects having fever in the last 24 hours. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 94 | 38 | 29 | 50 | 641
Days
  6M-4Y, DaFs: number analyzed (Participants) | 41 | 23 | 15 | 35 | 357
  6M-4Y, DaFs | 2.1 (1.35) | 2.7 (1.99) | 1.4 (0.51) | 2.0 (1.46) | 2.4 (1.76)
  5-19Y, DaFs: number analyzed (Participants) | 39 | 11 | 11 | 13 | 115
  5-19Y, DaFs | 2.5 (1.62) | 2.6 (2.38) | 2.5 (2.34) | 2.1 (1.80) | 2.1 (1.38)
  20+Y, DaFs: number analyzed (Participants) | 14 | 4 | 3 | 2 | 169
  20+Y, DaFs | 4.0 (3.64) | 2.0 (1.15) | 2.0 (1.00) | 4.0 (2.83) | 3.2 (2.96)

18. Secondary Outcome: Mean Number of Days With Fever at Survey 3
Description: The mean and standard deviation of the number of days ago with fever start (DaFs) were calculated for subjects having fever in the last 24 hours. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 134 | 72 | 36 | 62 | 619
Days
  6M-4Y, DaFs: number analyzed (Participants) | 60 | 44 | 28 | 44 | 360
  6M-4Y, DaFs | 2.3 (1.90) | 2.4 (1.95) | 2.2 (1.33) | 2.1 (1.37) | 2.5 (1.80)
  5-19Y, DaFs: number analyzed (Participants) | 54 | 24 | 4 | 17 | 92
  5-19Y, DaFs | 2.3 (1.58) | 2.8 (1.63) | 2.5 (1.73) | 1.8 (0.53) | 2.7 (2.21)
  20+Y, DaFs: number analyzed (Participants) | 20 | 4 | 4 | 1 | 167
  20+Y, DaFs | 3.0 (1.81) | 2.8 (0.50) | 3.8 (2.22) | 3.0 (0.00) | 3.3 (4.28)

19. Secondary Outcome: Mean Number of Days With Fever at Survey 4
Description: The mean and standard deviation of the number of days ago with fever start (DaFs) were calculated for subjects having fever in the last 24 hours. Fever data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: During the survey period (approximatively 1 year)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 88 | 26 | 9 | 31 | 162
Days
  6M-4Y, DaFs: number analyzed (Participants) | 39 | 18 | 5 | 27 | 115
  6M-4Y, DaFs | 2.2 (1.05) | 2.4 (2.43) | 1.6 (0.89) | 2.2 (1.64) | 2.7 (1.88)
  5-19Y, DaFs: number analyzed (Participants) | 38 | 8 | 4 | 4 | 22
  5-19Y, DaFs | 2.0 (0.97) | 3.8 (2.38) | 1.5 (0.58) | 2.0 (1.15) | 2.1 (1.23)
  20+Y, DaFs: number analyzed (Participants) | 11 | 0 | 0 | 0 | 25
  20+Y, DaFs | 2.5 (1.21) |  |  |  | 3.2 (1.38)

20. Secondary Outcome: Axillary Temperature at Visit in Survey 1
Description: The mean and standard deviation of the axillary temperature at visit (A temp. at V) were calculated. Axillary temperature data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 785 | 258 | 81 | 188 | 5087
Degrees Celsius
  6M-4Y, A temp. at V: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2479
  6M-4Y, A temp. at V | 36.65 (0.521) | 36.64 (0.623) | 36.72 (0.782) | 37.04 (0.803) | 36.55 (0.522)
  5-19Y, A temp. at V: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, A temp. at V | 36.56 (0.469) | 36.70 (0.597) | 37.07 (0.853) | 37.29 (0.928) | 36.63 (0.496)
  20+Y, A temp. at V: number analyzed (Participants) | 118 | 17 | 0 | 11 | 1441
  20+Y, A temp. at V | 36.55 (0.459) | 36.70 (0.387) |  | 36.82 (0.462) | 36.60 (0.478)

21. Secondary Outcome: Axillary Temperature at Visit in Survey 2
Description: The mean and standard deviation of axillary temperature at visit (A temp. at V) were calculated. Axillary temperature data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5221
Degrees Celsius
  6M-4Y, A temp. at V: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, A temp. at V | 36.69 (0.574) | 36.75 (0.628) | 36.86 (0.725) | 37.41 (1.201) | 36.60 (0.479)
  5-19Y, A temp. at V: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, A temp. at V | 36.70 (0.522) | 36.76 (0.507) | 36.76 (0.773) | 37.36 (0.949) | 36.66 (0.447)
  20+Y, A temp. at V: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1440
  20+Y, A temp. at V | 36.70 (0.478) | 36.75 (0.375) | 36.64 (0.559) | 37.09 (0.713) | 36.67 (0.430)

22. Secondary Outcome: Axillary Temperature at Visit in Survey 3
Description: The mean and standard deviation of axillary temperature at visit (A temp. at V) were calculated. Axillary temperature data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 267 | 92 | 130 | 5117
Degrees Celsius
  6M-4Y, A temp. at V: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, A temp. at V | 36.47 (0.517) | 36.66 (0.652) | 36.68 (0.701) | 36.97 (0.951) | 36.54 (0.496)
  5-19Y, A temp. at V: number analyzed (Participants) | 341 | 93 | 13 | 35 | 1128
  5-19Y, A temp. at V | 36.56 (0.551) | 36.66 (0.571) | 36.61 (0.475) | 37.45 (1.117) | 36.59 (0.462)
  20+Y, A temp. at V: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1401
  20+Y, A temp. at V | 36.44 (0.515) | 36.42 (0.409) | 37.54 (1.135) | 37.18 (0.727) | 36.55 (0.493)

23. Secondary Outcome: Axillary Temperature at Visit in Survey 4
Description: The mean and standard deviation of axillary temperature at visit (A temp. at V) were calculated. Axillary temperature data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1683
Degrees Celsius
  6M-4Y, A temp. at V: number analyzed (Participants) | 168 | 103 | 20 | 54 | 847
  6M-4Y, A temp. at V | 36.51 (0.508) | 36.51 (0.535) | 36.95 (0.927) | 37.16 (1.187) | 36.40 (0.492)
  5-19Y, A temp. at V: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, A temp. at V | 36.53 (0.510) | 36.55 (0.379) | 36.53 (0.570) | 36.61 (0.431) | 36.38 (0.430)
  20+Y, A temp. at V: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, A temp. at V | 36.42 (0.444) | 36.68 (0.206) |  | 36.50 (0.000) | 36.39 (0.457)

24. Secondary Outcome: Number of Subjects Living in the Same House at Survey 1
Description: The malaria prevention and risk factors characteristics were: Number of persons living in the same part of the house (PLSPH) among persons enrolled in the study (PES), in the following combinations: < y/x (less than [<] y PLSPH among x PES), y-z/x (y to z PLSPH among x PES), > z/x (more than [>] z PLSPH among x PES), y-z/> x (y to z PLSPH among more than [>] x PES), > z/> x (more than [>] z PLSPH among more than [>] x PES, or missing information). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, PLSPH/PES, <3/1: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, <3/1 | 34 | 13 | 3 | 2 | 78
  6M-4Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, 4-5/1 | 32 | 15 | 1 | 2 | 146
  6M-4Y, PLSPH/PES, >5/1: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, >5/1 | 20 | 10 | 0 | 3 | 123
  6M-4Y, PLSPH/PES, <3/2: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, <3/2 | 46 | 14 | 6 | 14 | 280
  6M-4Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, 4-5/2 | 106 | 49 | 13 | 36 | 737
  6M-4Y, PLSPH/PES, >5/2: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, >5/2 | 119 | 59 | 28 | 59 | 1038
  6M-4Y, PLSPH/PES, <3/3: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, <3/3 | 1 | 0 | 0 | 0 | 3
  6M-4Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, 4-5/3 | 1 | 1 | 1 | 1 | 19
  6M-4Y, PLSPH/PES, >5/3: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, >5/3 | 13 | 7 | 4 | 1 | 45
  6M-4Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 1 | 0 | 1
  6M-4Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PLSPH/PES, >5/>3 | 1 | 2 | 1 | 1 | 9
  6M-4Y, Missing: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, Missing | 0 | 0 | 0 | 0 | 1
  5-19Y, PLSPH/PES, <3/1: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, <3/1 | 20 | 6 | 0 | 0 | 28
  5-19Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, 4-5/1 | 14 | 2 | 1 | 1 | 17
  5-19Y, PLSPH/PES, >5/1: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, >5/1 | 8 | 3 | 1 | 0 | 37
  5-19Y, PLSPH/PES, <3/2: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, <3/2 | 19 | 4 | 1 | 5 | 75
  5-19Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, 4-5/2 | 76 | 13 | 9 | 17 | 357
  5-19Y, PLSPH/PES, >5/2: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, >5/2 | 111 | 38 | 10 | 34 | 560
  5-19Y, PLSPH/PES, <3/3: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, <3/3 | 0 | 1 | 0 | 0 | 2
  5-19Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, 4-5/3 | 10 | 1 | 0 | 0 | 14
  5-19Y, PLSPH/PES, >5/3: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, >5/3 | 25 | 2 | 1 | 1 | 59
  5-19Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, 4-5/>3 | 1 | 0 | 0 | 0 | 0
  5-19Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PLSPH/PES, >5/>3 | 10 | 1 | 0 | 0 | 17
  5-19Y, Missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, Missing | 0 | 0 | 0 | 0 | 1
  20+Y, PLSPH/PES, <3/1: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, <3/1 | 3 | 0 |  | 0 | 49
  20+Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, 4-5/1 | 1 | 0 |  | 0 | 16
  20+Y, PLSPH/PES, >5/1: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, >5/1 | 6 | 1 |  | 0 | 26
  20+Y, PLSPH/PES, <3/2: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, <3/2 | 22 | 2 |  | 2 | 234
  20+Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, 4-5/2 | 40 | 7 |  | 3 | 449
  20+Y, PLSPH/PES, >5/2: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, >5/2 | 33 | 7 |  | 6 | 575
  20+Y, PLSPH/PES, <3/3: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, <3/3 | 0 | 0 |  | 0 | 2
  20+Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, 4-5/3 | 3 | 0 |  | 0 | 18
  20+Y, PLSPH/PES, >5/3: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, >5/3 | 10 | 0 |  | 0 | 51
  20+Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, 4-5/>3 | 0 | 0 |  | 0 | 1
  20+Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PLSPH/PES, >5/>3 | 1 | 0 |  | 0 | 18
  20+Y, Missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, Missing | 0 | 0 |  | 0 | 2

25. Secondary Outcome: Number of Subjects Living in the Same House at Survey 2
Description: The malaria prevention and risk factors characteristics were: Number of persons living in the same part of the house (PLSPH) among persons enrolled in the study (PES), in the following combinations: < y/x (less than [<] y PLSPH among x PES), y-z/x (y to z PLSPH among x PES), > z/x (more than [>] z PLSPH among x PES), y-z/> x (y to z PLSPH among more than [>] x PES), > z/> x (more than [>] z PLSPH among more than [>] x PES, or missing information). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, PLSPH/PES, <3/1: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, <3/1 | 27 | 18 | 8 | 2 | 59
  6M-4Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, 4-5/1 | 33 | 18 | 8 | 3 | 112
  6M-4Y, PLSPH/PES, >5/1: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, >5/1 | 13 | 9 | 3 | 4 | 84
  6M-4Y, PLSPH/PES, <3/2: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, <3/2 | 37 | 21 | 8 | 14 | 306
  6M-4Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, 4-5/2 | 93 | 48 | 17 | 24 | 964
  6M-4Y, PLSPH/PES, >5/2: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, >5/2 | 76 | 32 | 19 | 27 | 1059
  6M-4Y, PLSPH/PES, <3/3: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, <3/3 | 1 | 0 | 0 | 0 | 2
  6M-4Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, 4-5/3 | 0 | 0 | 0 | 0 | 11
  6M-4Y, PLSPH/PES, >5/3: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, >5/3 | 3 | 1 | 4 | 2 | 24
  6M-4Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 2
  6M-4Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH/PES, >5/>3 | 0 | 1 | 0 | 0 | 0
  5-19Y, PLSPH/PES, <3/1: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, <3/1 | 34 | 3 | 1 | 3 | 23
  5-19Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, 4-5/1 | 30 | 13 | 2 | 0 | 20
  5-19Y, PLSPH/PES, >5/1: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, >5/1 | 16 | 3 | 0 | 0 | 38
  5-19Y, PLSPH/PES, <3/2: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, <3/2 | 30 | 3 | 0 | 2 | 69
  5-19Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, 4-5/2 | 98 | 17 | 10 | 13 | 426
  5-19Y, PLSPH/PES, >5/2: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, >5/2 | 105 | 28 | 15 | 17 | 548
  5-19Y, PLSPH/PES, <3/3: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, <3/3 | 2 | 0 | 0 | 0 | 1
  5-19Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, 4-5/3 | 4 | 0 | 0 | 0 | 9
  5-19Y, PLSPH/PES, >5/3: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, >5/3 | 14 | 4 | 1 | 1 | 20
  5-19Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 4
  5-19Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH/PES, >5/>3 | 0 | 0 | 0 | 0 | 0
  20+Y, PLSPH-PES, <3/1: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH-PES, <3/1 | 14 | 0 | 0 | 0 | 40
  20+Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, 4-5/1 | 8 | 0 | 0 | 0 | 26
  20+Y, PLSPH/PES, >5/1: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, >5/1 | 5 | 0 | 1 | 0 | 51
  20+Y, PLSPH/PES, <3/2: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, <3/2 | 34 | 2 | 1 | 2 | 253
  20+Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, 4-5/2 | 39 | 3 | 0 | 2 | 553
  20+Y, PLSPH/PES, >5/2: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, >5/2 | 21 | 5 | 3 | 3 | 476
  20+Y, PLSPH/PES, <3/3: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, <3/3 | 0 | 0 | 0 | 0 | 3
  20+Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, 4-5/3 | 0 | 0 | 0 | 0 | 9
  20+Y, PLSPH/PES, >5/3: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, >5/3 | 3 | 0 | 0 | 0 | 25
  20+Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 2
  20+Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH/PES, >5/>3 | 0 | 0 | 0 | 0 | 3

26. Secondary Outcome: Number of Subjects Living in the Same House at Survey 3
Description: The malaria prevention and risk factors characteristics were: Number of persons living in the same part of the house (PLSPH) among persons enrolled in the study (PES), in the following combinations: < y/x (less than [<] y PLSPH among x PES), y-z/x (y to z PLSPH among x PES), > z/x (more than [>] z PLSPH among x PES), y-z/> x (y to z PLSPH among more than [>] x PES), > z/> x (more than [>] z PLSPH among more than [>] x PES, or missing information). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, PLSPH/PES, <3/1: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, <3/1 | 31 | 16 | 7 | 11 | 63
  6M-4Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, 4-5/1 | 31 | 26 | 8 | 11 | 94
  6M-4Y, PLSPH/PES, >5/1: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, >5/1 | 15 | 10 | 6 | 2 | 94
  6M-4Y, PLSPH/PES, <3/2: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, <3/2 | 43 | 24 | 13 | 17 | 340
  6M-4Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, 4-5/2 | 76 | 30 | 19 | 22 | 973
  6M-4Y, PLSPH/PES, >5/2: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, >5/2 | 75 | 44 | 19 | 26 | 984
  6M-4Y, PLSPH/PES, <3/3: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, <3/3 | 0 | 0 | 0 | 0 | 0
  6M-4Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, 4-5/3 | 2 | 0 | 1 | 0 | 11
  6M-4Y, PLSPH/PES, >5/3: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, >5/3 | 6 | 11 | 1 | 2 | 29
  6M-4Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  6M-4Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH/PES, >5/>3 | 0 | 0 | 0 | 0 | 0
  5-19Y, PLSPH/PES, <3/1: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, <3/1 | 40 | 9 | 1 | 1 | 24
  5-19Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, 4-5/1 | 32 | 8 | 0 | 1 | 23
  5-19Y, PLSPH/PES, >5/1: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, >5/1 | 31 | 1 | 0 | 3 | 42
  5-19Y, PLSPH/PES, <3/2: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, <3/2 | 24 | 13 | 0 | 2 | 88
  5-19Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, 4-5/2 | 74 | 25 | 5 | 13 | 421
  5-19Y, PLSPH/PES, >5/2: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, >5/2 | 103 | 36 | 7 | 15 | 507
  5-19Y, PLSPH/PES, <3/3: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, <3/3 | 0 | 0 | 0 | 0 | 0
  5-19Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, 4-5/3 | 7 | 0 | 0 | 0 | 7
  5-19Y, PLSPH/PES, >5/3: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, >5/3 | 30 | 2 | 0 | 0 | 17
  5-19Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  5-19Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH/PES, >5/>3 | 0 | 0 | 0 | 0 | 0
  20+Y, PLSPH/PES, <3/1: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, <3/1 | 18 | 0 | 0 | 0 | 40
  20+Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, 4-5/1 | 7 | 0 | 0 | 0 | 27
  20+Y, PLSPH/PES, >5/1: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, >5/1 | 5 | 0 | 0 | 0 | 33
  20+Y, PLSPH/PES, <3/2: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, <3/2 | 43 | 3 | 0 | 1 | 273
  20+Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, 4-5/2 | 57 | 4 | 3 | 0 | 516
  20+Y, PLSPH/PES, >5/2: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, >5/2 | 28 | 6 | 2 | 3 | 463
  20+Y, PLSPH/PES, <3/3: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, <3/3 | 0 | 0 | 0 | 0 | 0
  20+Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, 4-5/3 | 0 | 0 | 0 | 0 | 14
  20+Y, PLSPH/PES, >5/3: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, >5/3 | 13 | 0 | 0 | 0 | 36
  20+Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  20+Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH/PES, >5/>3 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects Living in the Same House at Survey 4
Description: The malaria prevention and risk factors characteristics were: Number of persons living in the same part of the house (PLSPH) among persons enrolled in the study (PES), in the following combinations: < y/x (less than [<] y PLSPH among x PES), y-z/x (y to z PLSPH among x PES), > z/x (more than [>] z PLSPH among x PES), y-z/> x (y to z PLSPH among more than [>] x PES), > z/> x (more than [>] z PLSPH among more than [>] x PES, or missing information). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, PLSPH/PES, <3/1: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, <3/1 | 28 | 21 | 2 | 7 | 42
  6M-4Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, 4-5/1 | 24 | 14 | 4 | 5 | 74
  6M-4Y, PLSPH/PES, >5/1: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, >5/1 | 18 | 7 | 1 | 5 | 59
  6M-4Y, PLSPH/PES, <3/2: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, <3/2 | 27 | 18 | 3 | 10 | 74
  6M-4Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, 4-5/2 | 30 | 23 | 3 | 13 | 184
  6M-4Y, PLSPH/PES, >5/2: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, >5/2 | 25 | 12 | 4 | 12 | 338
  6M-4Y, PLSPH-PES, <3/3: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH-PES, <3/3 | 0 | 0 | 1 | 0 | 1
  6M-4Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, 4-5/3 | 1 | 1 | 0 | 1 | 9
  6M-4Y, PLSPH/PES, >5/3: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, >5/3 | 14 | 7 | 2 | 1 | 62
  6M-4Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 1
  6M-4Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH/PES, >5/>3 | 1 | 0 | 0 | 0 | 4
  5-19Y, PLSPH/PES, <3/1: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, <3/1 | 36 | 5 | 2 | 2 | 17
  5-19Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, 4-5/1 | 35 | 11 | 1 | 2 | 23
  5-19Y, PLSPH/PES, >5/1: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, >5/1 | 4 | 2 | 2 | 1 | 7
  5-19Y, PLSPH/PES, <3/2: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, <3/2 | 13 | 5 | 2 | 0 | 10
  5-19Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, 4-5/2 | 27 | 8 | 3 | 3 | 65
  5-19Y, PLSPH/PES, >5/2: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, >5/2 | 31 | 10 | 3 | 4 | 149
  5-19Y, PLSPH/PES, <3/3: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, <3/3 | 0 | 0 | 0 | 0 | 0
  5-19Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, 4-5/3 | 5 | 1 | 0 | 0 | 12
  5-19Y, PLSPH/PES, >5/3: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, >5/3 | 42 | 9 | 3 | 1 | 38
  5-19Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, 4-5/>3 | 0 | 0 | 0 | 0 | 2
  5-19Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH/PES, >5/>3 | 5 | 0 | 0 | 0 | 5
  20+Y, PLSPH/PES, <3/1: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, <3/1 | 4 | 0 |  | 0 | 20
  20+Y, PLSPH/PES, 4-5/1: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, 4-5/1 | 4 | 0 |  | 0 | 8
  20+Y, PLSPH/PES, >5/1: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, >5/1 | 1 | 0 |  | 0 | 10
  20+Y, PLSPH/PES, <3/2: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, <3/2 | 23 | 0 |  | 0 | 81
  20+Y, PLSPH/PES, 4-5/2: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, 4-5/2 | 26 | 2 |  | 0 | 119
  20+Y, PLSPH/PES, >5/2: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, >5/2 | 15 | 1 |  | 0 | 191
  20+Y, PLSPH/PES, <3/3: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, <3/3 | 1 | 0 |  | 0 | 3
  20+Y, PLSPH/PES, 4-5/3: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, 4-5/3 | 2 | 0 |  | 1 | 3
  20+Y, PLSPH/PES, >5/3: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, >5/3 | 11 | 1 |  | 0 | 67
  20+Y, PLSPH/PES, 4-5/>3: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, 4-5/>3 | 0 | 0 |  | 0 | 1
  20+Y, PLSPH/PES, >5/>3: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH/PES, >5/>3 | 0 | 0 |  | 0 | 5

28. Secondary Outcome: Mean Number of Subjects Living in the Same House at Survey 1
Description: The malaria prevention and risk factors characteristics were the following: the mean and standard deviation of the number of persons living in the same part of the house (PLSPH). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Persons
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Persons
  6M-4Y, PLSPH: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2479
  6M-4Y, PLSPH | 6.4 (4.83) | 6.3 (4.23) | 6.5 (3.98) | 5.8 (2.14) | 6.5 (4.28)
  5-19Y, PLSPH: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1166
  5-19Y, PLSPH | 6.9 (4.55) | 6.6 (3.53) | 5.9 (1.91) | 6.5 (3.04) | 7.1 (4.69)
  20+Y, PLSPH: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1439
  20+Y, PLSPH | 6.1 (4.15) | 7.4 (5.21) |  | 6.2 (2.99) | 6.3 (4.24)

29. Secondary Outcome: Mean Number of Subjects Living in the Same House at Survey 2
Description: The malaria prevention and risk factors characteristics were the following: the mean and standard deviation of the number of persons living in the same part of the house (PLSPH). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Persons
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Persons
  6M-4Y, PLSPH: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PLSPH | 5.1 (2.90) | 5.0 (2.17) | 5.1 (2.34) | 5.4 (2.62) | 5.8 (2.66)
  5-19Y, PLSPH: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PLSPH | 5.5 (2.64) | 6.1 (2.78) | 5.9 (1.89) | 5.9 (2.81) | 6.2 (2.78)
  20+Y, PLSPH: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PLSPH | 4.7 (3.35) | 6.5 (3.24) | 7.8 (3.27) | 5.3 (2.56) | 5.4 (2.64)

30. Secondary Outcome: Mean Number of Subjects Living in the Same House at Survey 3
Description: The malaria prevention and risk factors characteristics were the following: the mean and standard deviation of the number of persons living in the same part of the house (PLSPH). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Persons
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Persons
  6M-4Y, PLSPH: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PLSPH | 5.1 (2.73) | 5.4 (2.74) | 5.1 (3.40) | 5.0 (2.43) | 5.6 (2.48)
  5-19Y, PLSPH: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PLSPH | 5.9 (3.25) | 5.1 (2.04) | 5.5 (1.85) | 5.8 (2.06) | 6.0 (2.42)
  20+Y, PLSPH: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PLSPH | 4.5 (2.16) | 5.9 (3.23) | 5.4 (1.14) | 6.5 (2.89) | 5.4 (2.77)

31. Secondary Outcome: Mean Number of Subjects Living in the Same House at Survey 4
Description: The malaria prevention and risk factors characteristics were the following: the mean and standard deviation of the number of persons living in the same part of the house (PLSPH). Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Persons
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Persons
  6M-4Y, PLSPH: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, PLSPH | 5.4 (3.12) | 5.1 (3.73) | 5.5 (3.50) | 5.2 (3.24) | 6.6 (3.33)
  5-19Y, PLSPH: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PLSPH | 6.5 (4.55) | 6.1 (3.95) | 6.3 (3.13) | 6.8 (4.28) | 7.3 (3.70)
  20+Y, PLSPH: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PLSPH | 5.0 (2.94) | 6.3 (2.22) |  | 5.0 (0.00) | 6.6 (3.96)

32. Secondary Outcome: Number of Subjects by Localisation and Type of Location at Survey 1
Description: The malaria prevention and risk factors characteristics were the following: localisation categories (i.e.: rural, urban, semi-rural or missing) and Type of Location (i.e.: Large city: >1 million habitants; Small city: >50000 & < 1 million habitants; Town: > 10000 and < 50000 habitants; Countryside: < 10000 habitants or missing type of location).
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, rural: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, rural | 309 | 136 | 45 | 106 | 1415
  6M-4Y, urban: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, urban | 39 | 22 | 10 | 11 | 803
  6M-4Y, semi-rural: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, semi-rural | 25 | 12 | 3 | 2 | 262
  6M-4Y, missing - localisation: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, missing - localisation | 0 | 0 | 0 | 0 | 0
  6M-4Y, large city: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, large city | 18 | 14 | 7 | 7 | 355
  6M-4Y, small city: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, small city | 0 | 0 | 0 | 0 | 18
  6M-4Y, town: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, town | 44 | 16 | 5 | 6 | 644
  6M-4Y, countryside: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, countryside | 311 | 140 | 46 | 106 | 1463
  5-19Y, rural: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, rural | 225 | 55 | 16 | 51 | 688
  5-19Y, urban: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, urban | 50 | 13 | 4 | 5 | 350
  5-19Y, semi-rural: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, semi-rural | 19 | 3 | 3 | 2 | 128
  5-19Y, missing - localisation: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, missing - localisation | 0 | 0 | 0 | 0 | 1
  5-19Y, large city: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, large city | 25 | 5 | 4 | 4 | 162
  5-19Y, small city: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, small city | 1 | 0 | 0 | 0 | 7
  5-19Y, town: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, town | 43 | 11 | 2 | 3 | 282
  5-19Y, countryside: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, countryside | 225 | 55 | 17 | 51 | 715
  5-19Y, missing - type of localisation: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, missing - type of localisation | 0 | 0 | 0 | 0 | 1
  20+Y, rural: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, rural | 89 | 12 |  | 10 | 923
  20+Y, urban: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, urban | 26 | 3 |  | 0 | 370
  20+Y, semi-rural: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, semi-rural | 4 | 2 |  | 1 | 147
  20+Y, missing - localisation: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, missing - localisation | 0 | 0 |  | 0 | 1
  20+Y, large city: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, large city | 16 | 3 |  | 0 | 181
  20+Y, small city: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, small city | 0 | 0 |  | 0 | 9
  20+Y, town: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, town | 14 | 2 |  | 1 | 299
  20+Y, countryside: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, countryside | 89 | 12 |  | 10 | 951
  20+Y, missing - type of localisation: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, missing - type of localisation | 0 | 0 |  | 0 | 1

33. Secondary Outcome: Number of Subjects by Localisation and Type of Location at Survey 2
Description: The malaria prevention and risk factors characteristics were the following: localisation categories (i.e.: rural, urban, semi-rural) and Type of Location (i.e.: Large city: >1 million habitants; Small city: >50000 & < 1 million habitants; Town: > 10000 and < 50000 habitants; Countryside: < 10000 habitants).
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, rural: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, rural | 212 | 120 | 51 | 60 | 1377
  6M-4Y, urban: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, urban | 44 | 16 | 14 | 15 | 995
  6M-4Y, semi-rural: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, semi-rural | 27 | 12 | 2 | 1 | 251
  6M-4Y, large city: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, large city | 10 | 4 | 5 | 6 | 374
  6M-4Y, small city: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, small city | 0 | 0 | 0 | 0 | 6
  6M-4Y, town: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, town | 34 | 12 | 9 | 9 | 632
  6M-4Y, countryside: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, countryside | 239 | 132 | 53 | 61 | 1611
  5-19Y, rural: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, rural | 237 | 48 | 17 | 25 | 583
  5-19Y, urban: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, urban | 72 | 22 | 11 | 10 | 472
  5-19Y, semi-rural: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, semi-rural | 24 | 1 | 1 | 1 | 103
  5-19Y, large city: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, large city | 15 | 5 | 2 | 7 | 172
  5-19Y, small city: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, small city | 0 | 0 | 0 | 0 | 1
  5-19Y, town: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, town | 57 | 17 | 9 | 3 | 305
  5-19Y, countryside: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, countryside | 261 | 49 | 18 | 26 | 680
  20+Y, rural: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, rural | 94 | 6 | 2 | 6 | 769
  20+Y, urban: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, urban | 26 | 4 | 3 | 1 | 515
  20+Y, semi-rural: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, semi-rural | 4 | 0 | 0 | 0 | 157
  20+Y, large city: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, large city | 6 | 2 | 0 | 1 | 191
  20+Y, small city: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, small city | 0 | 0 | 0 | 0 | 5
  20+Y, town: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, town | 20 | 2 | 3 | 0 | 330
  20+Y, countryside: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, countryside | 98 | 6 | 2 | 6 | 915

34. Secondary Outcome: Number of Subjects by Localisation and Type of Location at Survey 3
Description: The malaria prevention and risk factors characteristics were the following: localisation categories (i.e.: rural, urban, semi-rural) and Type of Location (i.e.: Large city: >1 million habitants; Small city: >50000 & < 1 million habitants; Town: > 10000 and < 50000 habitants; Countryside: < 10000 habitants).
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, rural: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, rural | 234 | 146 | 65 | 82 | 1531
  6M-4Y, urban: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, urban | 30 | 11 | 5 | 5 | 881
  6M-4Y, semi-rural: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, semi-rural | 15 | 4 | 4 | 4 | 176
  6M-4Y, large city: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, large city | 7 | 3 | 1 | 3 | 386
  6M-4Y, small city: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, small city | 0 | 0 | 0 | 0 | 2
  6M-4Y, town: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, town | 23 | 9 | 4 | 2 | 541
  6M-4Y, countryside: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, countryside | 249 | 149 | 69 | 86 | 1659
  5-19Y, rural: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, rural | 283 | 78 | 9 | 28 | 645
  5-19Y, urban: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, urban | 42 | 12 | 4 | 7 | 404
  5-19Y, semi-rural: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, semi-rural | 16 | 4 | 0 | 0 | 80
  5-19Y, large city: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, large city | 12 | 2 | 2 | 2 | 182
  5-19Y, small city: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, small city | 0 | 0 | 0 | 0 | 1
  5-19Y, town: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, town | 30 | 10 | 2 | 5 | 241
  5-19Y, countryside: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, countryside | 299 | 82 | 9 | 28 | 705
  20+Y, rural: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, rural | 147 | 8 | 5 | 3 | 868
  20+Y, urban: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, urban | 23 | 3 | 0 | 1 | 430
  20+Y, semi-rural: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, semi-rural | 1 | 2 | 0 | 0 | 104
  20+Y, large city: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, large city | 15 | 0 | 0 | 0 | 185
  20+Y, small city: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, small city | 0 | 0 | 0 | 0 | 1
  20+Y, town: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, town | 8 | 3 | 0 | 1 | 273
  20+Y, countryside: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, countryside | 148 | 10 | 5 | 3 | 943

35. Secondary Outcome: Number of Subjects by Localisation and Type of Location at Survey 4
Description: The malaria prevention and risk factors characteristics were the following: localisation categories (i.e.: rural, urban, semi-rural) and Type of Location (i.e.: Large city: >1 million habitants; Small city: >50000 & < 1 million habitants; Town: > 10000 and < 50000 habitants; Countryside: < 10000 habitants).
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, rural: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, rural | 153 | 102 | 20 | 53 | 536
  6M-4Y, urban: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, urban | 15 | 1 | 0 | 1 | 312
  6M-4Y, semi-rural: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, semi-rural | 0 | 0 | 0 | 0 | 0
  6M-4Y, large city: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, large city | 0 | 0 | 0 | 0 | 0
  6M-4Y, small city: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, small city | 0 | 0 | 0 | 0 | 0
  6M-4Y, town: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, town | 15 | 1 | 0 | 1 | 311
  6M-4Y, countryside: number analyzed (Participants) | 168 | 103 | 20 | 54 | 848
  6M-4Y, countryside | 153 | 102 | 20 | 53 | 537
  5-19Y, rural: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, rural | 184 | 49 | 14 | 11 | 186
  5-19Y, urban: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, urban | 14 | 2 | 2 | 2 | 142
  5-19Y, semi-rural: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, semi-rural | 0 | 0 | 0 | 0 | 0
  5-19Y, large city: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, large city | 0 | 0 | 0 | 0 | 0
  5-19Y, small city: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, small city | 0 | 0 | 0 | 0 | 0
  5-19Y, town: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, town | 14 | 2 | 2 | 2 | 141
  5-19Y, countryside: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, countryside | 184 | 49 | 14 | 11 | 187
  20+Y, rural: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, rural | 85 | 4 |  | 1 | 352
  20+Y, urban: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, urban | 2 | 0 |  | 0 | 156
  20+Y, semi-rural: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, semi-rural | 0 | 0 |  | 0 | 0
  20+Y, large city: number analyzed (Participants) | 453 | 4 | 0 | 1 | 508
  20+Y, large city | 0 | 0 |  | 0 | 0
  20+Y, small city: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, small city | 0 | 0 |  | 0 | 0
  20+Y, town: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, town | 2 | 0 |  | 0 | 155
  20+Y, countryside: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, countryside | 85 | 4 |  | 1 | 353

36. Secondary Outcome: Number of Subjects by House Construction Material Regarding Walls and Floor at Survey 1
Description: The malaria prevention and risk factors characteristics were the following: Main house construction material (MHCM) walls and MHCM floor. MHCM walls data were assessed for the following sub-categories: mud, brick, cement/plaster, cement/paint, other and missing. MHCM floor data were assessed for the following sub-categories: natural floor, rudimentary floor, parquet polished wood, vinyl or asphalt strips, ceramic tiles, cement, carpet, missing. Note: Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, MHCM walls - mud: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM walls - mud | 97 | 62 | 34 | 84 | 869
  6M-4Y, MHCM walls - brick: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM walls - brick | 190 | 76 | 12 | 12 | 504
  6M-4Y, MHCM walls - cement/plaster: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM walls - cement/plaster | 41 | 16 | 7 | 11 | 383
  6M-4Y, MHCM walls - cement/paint: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM walls - cement/paint | 29 | 12 | 5 | 11 | 408
  6M-4Y, MHCM walls - other: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM walls - other | 16 | 4 | 0 | 1 | 316
  6M-4Y, MHCM floor - natural floor: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - natural floor | 197 | 100 | 42 | 83 | 1079
  6M-4Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 3
  6M-4Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - parquet polished wood | 0 | 0 | 0 | 0 | 2
  6M-4Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 4
  6M-4Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - ceramic tiles | 0 | 1 | 0 | 0 | 30
  6M-4Y, MHCM floor - cement: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - cement | 170 | 69 | 16 | 33 | 1309
  6M-4Y, MHCM floor - carpet: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM floor - carpet | 6 | 0 | 0 | 3 | 53
  5-19Y, MHCM walls - mud: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - mud | 89 | 29 | 13 | 48 | 424
  5-19Y, MHCM walls - brick: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - brick | 119 | 23 | 3 | 4 | 223
  5-19Y, MHCM walls - cement/plaster: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - cement/plaster | 43 | 8 | 4 | 5 | 168
  5-19Y, MHCM walls - cement/paint: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - cement/paint | 30 | 4 | 3 | 1 | 186
  5-19Y, MHCM walls - other: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - other | 13 | 7 | 0 | 0 | 165
  5-19Y, MHCM walls - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM walls - missing | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM floor - natural floor: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - natural floor | 146 | 46 | 12 | 48 | 511
  5-19Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - parquet polished wood | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 2
  5-19Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - ceramic tiles | 0 | 1 | 0 | 0 | 14
  5-19Y, MHCM floor - cement: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - cement | 146 | 24 | 11 | 10 | 607
  5-19Y, MHCM floor - carpet: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - carpet | 2 | 0 | 0 | 0 | 30
  5-19Y, MHCM floor - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM floor - missing | 0 | 0 | 0 | 0 | 1
  20+Y, MHCM walls - mud: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - mud | 43 | 7 |  | 9 | 548
  20+Y, MHCM walls - brick: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - brick | 43 | 2 |  | 0 | 337
  20+Y, MHCM walls - cement/plaster: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - cement/plaster | 12 | 5 |  | 1 | 192
  20+Y, MHCM walls - cement/paint: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - cement/paint | 16 | 3 |  | 0 | 217
  20+Y, MHCM walls - other: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - other | 5 | 0 |  | 1 | 146
  20+Y, MHCM walls - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM walls - missing | 0 | 0 |  | 0 | 1
  20+Y, MHCM floor - natural floor: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - natural floor | 64 | 5 |  | 8 | 690
  20+Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - rudimentary floor | 0 | 0 |  | 0 | 2
  20+Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - parquet polished wood | 0 | 0 |  | 0 | 1
  20+Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - vinyl/asphalt strips | 0 | 0 |  | 0 | 2
  20+Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - ceramic tiles | 0 | 0 |  | 0 | 13
  20+Y, MHCM floor - cement: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - cement | 55 | 11 |  | 3 | 705
  20+Y, MHCM floor - carpet: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - carpet | 0 | 1 |  | 0 | 27
  20+Y, MHCM floor - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM floor - missing | 0 | 0 |  | 0 | 1

37. Secondary Outcome: Number of Subjects by House Construction Material Regarding Walls and Floor at Survey 2
Description: The malaria prevention and risk factors characteristics were the following: Main house construction material (MHCM) walls and MHCM floor. MHCM walls data were assessed for the following sub-categories: mud, brick, cement/plaster, cement/paint, other. MHCM floor data were assessed for the following sub-categories: natural floor, rudimentary floor, parquet polished wood, vinyl or asphalt strips, ceramic tiles, cement, carpet. Note: Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, MHCM walls - mud: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM walls - mud | 49 | 30 | 15 | 29 | 1010
  6M-4Y, MHCM walls - brick: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM walls - brick | 163 | 81 | 34 | 31 | 458
  6M-4Y, MHCM walls - cement/plaster: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM walls - cement/plaster | 33 | 14 | 8 | 8 | 472
  6M-4Y, MHCM walls - cement/paint: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM walls - cement/paint | 32 | 15 | 4 | 2 | 393
  6M-4Y, MHCM walls - other: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM walls - other | 6 | 8 | 6 | 6 | 290
  6M-4Y, MHCM floor - natural floor: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - natural floor | 194 | 97 | 45 | 53 | 1145
  6M-4Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 2
  6M-4Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - parquet polished wood | 0 | 0 | 1 | 0 | 6
  6M-4Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 15
  6M-4Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - ceramic tiles | 0 | 1 | 0 | 1 | 40
  6M-4Y, MHCM floor - cement: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - cement | 84 | 50 | 20 | 22 | 1357
  6M-4Y, MHCM floor - carpet: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM floor - carpet | 5 | 0 | 1 | 0 | 58
  5-19Y, MHCM walls - mud: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM walls - mud | 79 | 20 | 11 | 21 | 445
  5-19Y, MHCM walls - brick: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM walls - brick | 155 | 26 | 11 | 7 | 191
  5-19Y, MHCM walls - cement/plaster: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM walls - cement/plaster | 51 | 15 | 2 | 4 | 207
  5-19Y, MHCM walls - cement/paint: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM walls - cement/paint | 34 | 5 | 1 | 0 | 182
  5-19Y, MHCM walls - other: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM walls - other | 14 | 5 | 4 | 4 | 133
  5-19Y, MHCM floor - natural floor: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - natural floor | 207 | 42 | 17 | 26 | 508
  5-19Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - rudimentary floor | 1 | 0 | 0 | 0 | 0
  5-19Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - parquet polished wood | 0 | 0 | 1 | 0 | 5
  5-19Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 10
  5-19Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - ceramic tiles | 0 | 0 | 0 | 0 | 26
  5-19Y, MHCM floor - cement: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - cement | 117 | 29 | 11 | 9 | 587
  5-19Y, MHCM floor - carpet: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM floor - carpet | 8 | 0 | 0 | 1 | 22
  20+Y, MHCM walls - mud: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM walls - mud | 26 | 5 | 1 | 5 | 520
  20+Y, MHCM walls - brick: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM walls - brick | 69 | 2 | 0 | 0 | 302
  20+Y, MHCM walls - cement/plaster: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM walls - cement/plaster | 7 | 0 | 1 | 1 | 258
  20+Y, MHCM walls - cement/paint: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM walls - cement/paint | 15 | 0 | 0 | 0 | 215
  20+Y, MHCM walls - other: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM walls - other | 7 | 3 | 3 | 1 | 146
  20+Y, MHCM floor - natural floor: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - natural floor | 88 | 7 | 2 | 5 | 653
  20+Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 1
  20+Y, MHCM floor - parquet polished wood: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - parquet polished wood | 0 | 0 | 0 | 0 | 1
  20+Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 1 | 0 | 4
  20+Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - ceramic tiles | 1 | 0 | 0 | 0 | 15
  20+Y, MHCM floor - cement: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - cement | 34 | 3 | 2 | 2 | 732
  20+Y, MHCM floor - carpet: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM floor - carpet | 1 | 0 | 0 | 0 | 35

38. Secondary Outcome: Number of Subjects by House Construction Material Regarding Walls and Floor at Survey 3
Description: The malaria prevention and risk factors characteristics were the following: Main house construction material (MHCM) walls and MHCM floor. MHCM walls data were assessed for the following sub-categories: mud, brick, cement/plaster, cement/paint, other. MHCM floor data were assessed for the following sub-categories: natural floor, rudimentary floor, ceramic tiles, cement, carpet. Note: Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo. Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, MHCM walls - mud: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM walls - mud | 65 | 42 | 19 | 33 | 969
  6M-4Y, MHCM walls - brick: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM walls - brick | 143 | 91 | 41 | 43 | 485
  6M-4Y, MHCM walls - cement/plaster: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM walls - cement/plaster | 23 | 10 | 10 | 5 | 350
  6M-4Y, MHCM walls - cement/paint: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM walls - cement/paint | 28 | 12 | 3 | 5 | 464
  6M-4Y, MHCM walls - other: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM walls - other | 20 | 6 | 1 | 5 | 320
  6M-4Y, MHCM floor - natural floor: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM floor - natural floor | 188 | 111 | 54 | 65 | 1082
  6M-4Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 4
  6M-4Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM floor - ceramic tiles | 1 | 0 | 0 | 0 | 26
  6M-4Y, MHCM floor - cement: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM floor - cement | 85 | 49 | 20 | 25 | 1406
  6M-4Y, MHCM floor - carpet: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM floor - carpet | 5 | 1 | 0 | 1 | 70
  5-19Y, MHCM walls - mud: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM walls - mud | 90 | 32 | 4 | 13 | 432
  5-19Y, MHCM walls - brick: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM walls - brick | 161 | 42 | 2 | 12 | 205
  5-19Y, MHCM walls - cement/plaster: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM walls - cement/plaster | 38 | 8 | 1 | 3 | 136
  5-19Y, MHCM walls - cement/paint: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM walls - cement/paint | 41 | 5 | 2 | 2 | 214
  5-19Y, MHCM walls - other: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM walls - other | 11 | 7 | 4 | 5 | 142
  5-19Y, MHCM floor - natural floor: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM floor - natural floor | 185 | 67 | 7 | 24 | 449
  5-19Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM floor - rudimentary floor | 0 | 1 | 0 | 0 | 0
  5-19Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM floor - ceramic tiles | 2 | 0 | 0 | 0 | 12
  5-19Y, MHCM floor - cement: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM floor - cement | 149 | 26 | 6 | 11 | 636
  5-19Y, MHCM floor - carpet: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM floor - carpet | 5 | 0 | 0 | 0 | 32
  20+Y, MHCM walls - mud: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM walls - mud | 46 | 3 | 4 | 3 | 520
  20+Y, MHCM walls - brick: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM walls - brick | 90 | 4 | 0 | 0 | 298
  20+Y, MHCM walls - cement/plaster: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM walls - cement/plaster | 10 | 0 | 1 | 0 | 188
  20+Y, MHCM walls - cement/paint: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM walls - cement/paint | 15 | 1 | 0 | 0 | 228
  20+Y, MHCM walls - other: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM walls - other | 10 | 5 | 0 | 1 | 168
  20+Y, MHCM floor - natural floor: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM floor - natural floor | 124 | 9 | 4 | 3 | 651
  20+Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 2
  20+Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM floor - ceramic tiles | 0 | 1 | 0 | 0 | 12
  20+Y, MHCM floor - cement: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM floor - cement | 46 | 3 | 1 | 1 | 699
  20+Y, MHCM floor - carpet: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM floor - carpet | 1 | 0 | 0 | 0 | 38

39. Secondary Outcome: Number of Subjects by House Construction Material Regarding Walls and Floor at Survey 4
Description: The malaria prevention and risk factors characteristics were the following: Main house construction material (MHCM) walls and MHCM floor. MHCM walls data were assessed for the following sub-categories: mud, brick, cement/plaster, cement/paint, other. MHCM floor data were assessed for the following sub-categories: natural floor, rudimentary floor, vinyl or asphalt strips, ceramic tiles, cement, carpet. Note: Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, MHCM walls - mud: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM walls - mud | 33 | 14 | 2 | 14 | 127
  6M-4Y, MHCM walls - brick: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM walls - brick | 92 | 76 | 17 | 33 | 231
  6M-4Y, MHCM walls - cement/plaster: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM walls - cement/plaster | 23 | 8 | 1 | 2 | 120
  6M-4Y, MHCM walls - cement/paint: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM walls - cement/paint | 6 | 2 | 0 | 1 | 81
  6M-4Y, MHCM walls - other: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM walls - other | 14 | 3 | 0 | 4 | 289
  6M-4Y, MHCM floor - natural floor: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - natural floor | 97 | 76 | 15 | 37 | 267
  6M-4Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - rudimentary floor | 0 | 1 | 0 | 0 | 0
  6M-4Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 2
  6M-4Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - ceramic tiles | 0 | 1 | 0 | 0 | 16
  6M-4Y, MHCM floor - cement: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - cement | 70 | 23 | 5 | 16 | 541
  6M-4Y, MHCM floor - carpet: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM floor - carpet | 1 | 2 | 0 | 1 | 22
  5-19Y, MHCM walls - mud: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM walls - mud | 40 | 4 | 0 | 2 | 36
  5-19Y, MHCM walls - brick: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM walls - brick | 114 | 27 | 9 | 5 | 78
  5-19Y, MHCM walls - cement/plaster: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM walls - cement/plaster | 24 | 11 | 4 | 1 | 52
  5-19Y, MHCM walls - cement/paint: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM walls - cement/paint | 13 | 4 | 1 | 0 | 30
  5-19Y, MHCM walls - other: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM walls - other | 7 | 5 | 2 | 5 | 132
  5-19Y, MHCM floor - natural floor: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - natural floor | 105 | 27 | 9 | 6 | 96
  5-19Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - rudimentary floor | 0 | 0 | 0 | 0 | 0
  5-19Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - vinyl/asphalt strips | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - ceramic tiles | 0 | 0 | 0 | 0 | 9
  5-19Y, MHCM floor - cement: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - cement | 89 | 24 | 7 | 7 | 214
  5-19Y, MHCM floor - carpet: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM floor - carpet | 4 | 0 | 0 | 0 | 8
  20+Y, MHCM walls - mud: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM walls - mud | 18 | 0 |  | 1 | 76
  20+Y, MHCM walls - brick: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM walls - brick | 52 | 1 |  | 0 | 171
  20+Y, MHCM walls - cement/plaster: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM walls - cement/plaster | 13 | 2 |  | 0 | 70
  20+Y, MHCM walls - cement/paint: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM walls - cement/paint | 1 | 0 |  | 0 | 38
  20+Y, MHCM walls - other: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM walls - other | 3 | 1 |  | 0 | 153
  20+Y, MHCM floor - natural floor: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - natural floor | 50 | 1 |  | 0 | 201
  20+Y, MHCM floor - rudimentary floor: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - rudimentary floor | 0 | 0 |  | 0 | 1
  20+Y, MHCM floor - vinyl/asphalt strips: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - vinyl/asphalt strips | 0 | 0 |  | 0 | 1
  20+Y, MHCM floor - ceramic tiles: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - ceramic tiles | 0 | 0 |  | 0 | 8
  20+Y, MHCM floor - cement: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - cement | 37 | 3 |  | 1 | 287
  20+Y, MHCM floor - carpet: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM floor - carpet | 0 | 0 |  | 0 | 10

40. Secondary Outcome: Number of Subjects Classified by House Construction Material Regarding Roof, Window/Eaves and Nets at Survey 1
Description: The malaria prevention and risk factors characteristics were the following: main house construction material (MHCM) roof, windows/eaves, nets. MHCM roof data were assessed for the following sub-categories: grass/palm, iron sheet, tiles, other, missing. MHCM windows/eaves data were assessed for the following sub-categories: closed, open, partially open, missing. MHCM nets data were assessed for the following sub-categories: nets not present, nets present on all windows, nets present on some windows, missing.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, MHCM roof - grass/palm: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM roof - grass/palm | 112 | 53 | 22 | 44 | 453
  6M-4Y, MHCM roof - iron sheet: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM roof - iron sheet | 231 | 109 | 35 | 74 | 1980
  6M-4Y, MHCM roof - tiles: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 7
  6M-4Y, MHCM roof - other: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM roof - other | 30 | 8 | 1 | 1 | 40
  6M-4Y, MHCM windows/eaves - closed: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM windows/eaves - closed | 193 | 93 | 31 | 77 | 1467
  6M-4Y, MHCM windows/eaves - open: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM windows/eaves - open | 76 | 33 | 17 | 20 | 486
  6M-4Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM windows/eaves - partially open | 104 | 44 | 10 | 22 | 527
  6M-4Y, MHCM windows/eaves - missing: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM windows/eaves - missing | 0 | 0 | 0 | 0 | 0
  6M-4Y, MHCM, nets - not present: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM, nets - not present | 322 | 157 | 54 | 91 | 1795
  6M-4Y, MHCM, nets - present on all windows: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM, nets - present on all windows | 26 | 6 | 1 | 21 | 450
  6M-4Y, MHCM, nets - present on some windows: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MHCM, nets - present on some windows | 25 | 7 | 3 | 7 | 235
  5-19Y, MHCM roof - grass/palm: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM roof - grass/palm | 88 | 19 | 7 | 28 | 212
  5-19Y, MHCM roof - iron sheet: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM roof - iron sheet | 193 | 48 | 16 | 30 | 944
  5-19Y, MHCM roof - tiles: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 2
  5-19Y, MHCM roof - other: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM roof - other | 13 | 4 | 0 | 0 | 8
  5-19Y, MHCM roof - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM roof - missing | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM windows/eaves - closed: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM windows/eaves - closed | 154 | 44 | 14 | 38 | 669
  5-19Y, MHCM windows/eaves - open: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM windows/eaves - open | 71 | 16 | 5 | 9 | 233
  5-19Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM windows/eaves - partially open | 69 | 11 | 4 | 11 | 264
  5-19Y, MHCM windows/eaves - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM windows/eaves - missing | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM, nets - not present: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM, nets - not present | 256 | 63 | 21 | 42 | 853
  5-19Y, MHCM, nets - present on all windows: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM, nets - present on all windows | 22 | 6 | 1 | 11 | 197
  5-19Y, MHCM, nets - present on some windows: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM, nets - present on some windows | 16 | 2 | 1 | 5 | 116
  5-19Y, MHCM, nets - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MHCM, nets - missing | 0 | 0 | 0 | 0 | 1
  20+Y, MHCM roof - grass/palm: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM roof - grass/palm | 31 | 5 |  | 3 | 280
  20+Y, MHCM roof - iron sheet: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM roof - iron sheet | 84 | 12 |  | 8 | 1117
  20+Y, MHCM roof - tiles: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM roof - tiles | 0 | 0 |  | 0 | 6
  20+Y, MHCM roof - other: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM roof - other | 4 | 0 |  | 0 | 37
  20+Y, MHCM roof - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM roof - missing | 0 | 0 |  | 0 | 1
  20+Y, MHCM windows/eaves - closed: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM windows/eaves - closed | 65 | 8 |  | 5 | 798
  20+Y, MHCM windows/eaves - open: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM windows/eaves - open | 25 | 5 |  | 2 | 291
  20+Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM windows/eaves - partially open | 29 | 4 |  | 4 | 351
  20+Y, MHCM windows/eaves - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM windows/eaves - missing | 0 | 0 |  | 0 | 1
  20+Y, MHCM, nets - not present: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM, nets - not present | 107 | 12 |  | 7 | 1081
  20+Y, MHCM, nets - present on all windows: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM, nets - present on all windows | 8 | 3 |  | 2 | 223
  20+Y, MHCM, nets - present on some windows: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM, nets - present on some windows | 4 | 2 |  | 2 | 136
  20+Y, MHCM, nets - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MHCM, nets - missing | 0 | 0 |  | 0 | 1

41. Secondary Outcome: Number of Subjects Classified by House Construction Material Regarding Roof, Window/Eaves and Nets at Survey 2
Description: The malaria prevention and risk factors characteristics were the following: main house construction material (MHCM) roof, windows/eaves, nets. MHCM roof data were assessed for the following sub-categories: grass/palm, iron sheet, tiles, other. MHCM windows/eaves data were assessed for the following sub-categories: closed, open, partially open. MHCM nets data were assessed for the following sub-categories: nets not present, nets present on all windows, nets present on some windows.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, MHCM roof - grass/palm: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM roof - grass/palm | 52 | 32 | 16 | 23 | 509
  6M-4Y, MHCM roof - iron sheet: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM roof - iron sheet | 201 | 102 | 46 | 50 | 2092
  6M-4Y, MHCM roof - tiles: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 1
  6M-4Y, MHCM roof - other: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM roof - other | 30 | 14 | 5 | 3 | 21
  6M-4Y, MHCM windows/eaves - closed: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM windows/eaves - closed | 97 | 54 | 30 | 39 | 1411
  6M-4Y, MHCM windows/eaves - open: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM windows/eaves - open | 88 | 45 | 20 | 19 | 669
  6M-4Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM windows/eaves - partially open | 98 | 49 | 17 | 18 | 543
  6M-4Y, MHCM, nets - not present: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM, nets - not present | 242 | 136 | 62 | 66 | 1843
  6M-4Y, MHCM, nets - present on all windows: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM, nets - present on all windows | 26 | 6 | 4 | 8 | 626
  6M-4Y, MHCM, nets - present on some windows: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MHCM, nets - present on some windows | 15 | 6 | 1 | 2 | 154
  5-19Y, MHCM roof - grass/palm: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM roof - grass/palm | 76 | 15 | 3 | 13 | 207
  5-19Y, MHCM roof - iron sheet: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM roof - iron sheet | 241 | 54 | 26 | 23 | 940
  5-19Y, MHCM roof - tiles: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 0
  5-19Y, MHCM roof - other: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM roof - other | 16 | 2 | 0 | 0 | 11
  5-19Y, MHCM windows/eaves - closed: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM windows/eaves - closed | 159 | 36 | 16 | 14 | 610
  5-19Y, MHCM windows/eaves - open: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM windows/eaves - open | 85 | 24 | 6 | 17 | 294
  5-19Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM windows/eaves - partially open | 89 | 11 | 7 | 5 | 254
  5-19Y, MHCM, nets - not present: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM, nets - not present | 290 | 65 | 23 | 28 | 793
  5-19Y, MHCM, nets - present on all windows: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM, nets - present on all windows | 36 | 5 | 3 | 6 | 296
  5-19Y, MHCM, nets - present on some windows: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MHCM, nets - present on some windows | 7 | 1 | 3 | 2 | 69
  20+Y, MHCM roof - grass/palm: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM roof - grass/palm | 30 | 3 | 1 | 2 | 276
  20+Y, MHCM roof - iron sheet: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM roof - iron sheet | 80 | 7 | 4 | 5 | 1144
  20+Y, MHCM roof - tiles: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM roof - tiles | 1 | 0 | 0 | 0 | 2
  20+Y, MHCM roof - other: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM roof - other | 13 | 0 | 0 | 0 | 19
  20+Y, MHCM windows/eaves - closed: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM windows/eaves - closed | 49 | 6 | 3 | 4 | 732
  20+Y, MHCM windows/eaves - open: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM windows/eaves - open | 42 | 3 | 2 | 2 | 372
  20+Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM windows/eaves - partially open | 33 | 1 | 0 | 1 | 337
  20+Y, MHCM, nets - not present: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM, nets - not present | 115 | 9 | 3 | 4 | 1033
  20+Y, MHCM, nets - present on all windows: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM, nets - present on all windows | 5 | 0 | 2 | 3 | 320
  20+Y, MHCM, nets - present on some windows: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MHCM, nets - present on some windows | 4 | 1 | 0 | 0 | 88

42. Secondary Outcome: Number of Subjects Classified by House Construction Material Regarding Roof, Window/Eaves and Nets at Survey 3
Description: The malaria prevention and risk factors characteristics were the following: main house construction material (MHCM) roof, windows/eaves, nets. MHCM roof data were assessed for the following sub-categories: grass/palm, iron sheet, tiles, other. MHCM windows/eaves data were assessed for the following sub-categories: closed, open, partially open. MHCM nets data were assessed for the following sub-categories: nets not present, nets present on all windows, nets present on some windows.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, MHCM roof - grass/palm: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM roof - grass/palm | 55 | 35 | 12 | 26 | 464
  6M-4Y, MHCM roof - iron sheet: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM roof - iron sheet | 214 | 125 | 60 | 63 | 2111
  6M-4Y, MHCM roof - tiles: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM roof - tiles | 0 | 0 | 0 | 1 | 9
  6M-4Y, MHCM roof - other: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM roof - other | 10 | 1 | 2 | 1 | 4
  6M-4Y, MHCM windows/eaves - closed: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM windows/eaves - closed | 164 | 82 | 38 | 57 | 1352
  6M-4Y, MHCM windows/eaves - open: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM windows/eaves - open | 86 | 67 | 28 | 30 | 845
  6M-4Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM windows/eaves - partially open | 29 | 12 | 8 | 4 | 391
  6M-4Y, MHCM, nets - not present: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM, nets - not present | 244 | 149 | 63 | 84 | 1918
  6M-4Y, MHCM, nets - present on all windows: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM, nets - present on all windows | 21 | 10 | 6 | 4 | 532
  6M-4Y, MHCM, nets - present on some windows: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MHCM, nets - present on some windows | 14 | 2 | 5 | 3 | 138
  5-19Y, MHCM roof - grass/palm: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM roof - grass/palm | 76 | 16 | 1 | 5 | 186
  5-19Y, MHCM roof - iron sheet: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM roof - iron sheet | 264 | 77 | 12 | 30 | 940
  5-19Y, MHCM roof - tiles: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 1
  5-19Y, MHCM roof - other: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM roof - other | 1 | 1 | 0 | 0 | 2
  5-19Y, MHCM windows/eaves - closed: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM windows/eaves - closed | 165 | 58 | 9 | 18 | 593
  5-19Y, MHCM windows/eaves - open: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM windows/eaves - open | 143 | 26 | 2 | 16 | 357
  5-19Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM windows/eaves - partially open | 33 | 10 | 2 | 1 | 179
  5-19Y, MHCM, nets - not present: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM, nets - not present | 290 | 83 | 13 | 28 | 818
  5-19Y, MHCM, nets - present on all windows: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM, nets - present on all windows | 31 | 9 | 0 | 4 | 261
  5-19Y, MHCM, nets - present on some windows: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MHCM, nets - present on some windows | 20 | 2 | 0 | 3 | 50
  20+Y, MHCM roof - grass/palm: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM roof - grass/palm | 45 | 1 | 2 | 2 | 259
  20+Y, MHCM roof - iron sheet: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM roof - iron sheet | 123 | 12 | 3 | 2 | 1123
  20+Y, MHCM roof - tiles: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM roof - tiles | 0 | 0 | 0 | 0 | 9
  20+Y, MHCM roof - other: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM roof - other | 3 | 0 | 0 | 0 | 11
  20+Y, MHCM windows/eaves - closed: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM windows/eaves - closed | 112 | 9 | 4 | 1 | 715
  20+Y, MHCM windows/eaves - open: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM windows/eaves - open | 49 | 2 | 1 | 3 | 483
  20+Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM windows/eaves - partially open | 10 | 2 | 0 | 0 | 204
  20+Y, MHCM, nets - not present: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM, nets - not present | 153 | 12 | 4 | 4 | 1052
  20+Y, MHCM, nets - present on all windows: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM, nets - present on all windows | 11 | 0 | 0 | 0 | 262
  20+Y, MHCM, nets - present on some windows: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MHCM, nets - present on some windows | 7 | 1 | 1 | 0 | 88

43. Secondary Outcome: Number of Subjects Classified by House Construction Material Regarding Roof, Window/Eaves and Nets at Survey 4
Description: The malaria prevention and risk factors characteristics were the following: main house construction material (MHCM) roof, windows/eaves, nets. MHCM roof data were assessed for the following sub-categories: grass/palm, iron sheet, other. MHCM windows/eaves data were assessed for the following sub-categories: closed, open, partially open. MHCM nets data were assessed for the following sub-categories: nets not present, nets present on all windows, nets present on some windows.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, MHCM roof - grass/palm: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM roof - grass/palm | 51 | 29 | 6 | 17 | 161
  6M-4Y, MHCM roof - iron sheet: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM roof - iron sheet | 111 | 67 | 14 | 28 | 673
  6M-4Y, MHCM roof - other: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM roof - other | 6 | 7 | 0 | 9 | 14
  6M-4Y, MHCM windows/eaves - closed: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM windows/eaves - closed | 124 | 58 | 13 | 34 | 725
  6M-4Y, MHCM windows/eaves - open: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM windows/eaves - open | 15 | 13 | 1 | 5 | 66
  6M-4Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM windows/eaves - partially open | 29 | 32 | 6 | 15 | 57
  6M-4Y, MHCM, nets - not present: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM, nets - not present | 156 | 95 | 16 | 51 | 712
  6M-4Y, MHCM, nets - present on all windows: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM, nets - present on all windows | 8 | 1 | 2 | 2 | 79
  6M-4Y, MHCM, nets - present on some windows: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MHCM, nets - present on some windows | 4 | 7 | 2 | 1 | 57
  5-19Y, MHCM roof - grass/palm: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM roof - grass/palm | 55 | 10 | 1 | 2 | 51
  5-19Y, MHCM roof - iron sheet: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM roof - iron sheet | 134 | 37 | 13 | 9 | 276
  5-19Y, MHCM roof - other: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM roof - other | 9 | 4 | 2 | 2 | 1
  5-19Y, MHCM windows/eaves - closed: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM windows/eaves - closed | 139 | 32 | 11 | 9 | 292
  5-19Y, MHCM windows/eaves - open: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM windows/eaves - open | 24 | 8 | 4 | 1 | 17
  5-19Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM windows/eaves - partially open | 35 | 11 | 1 | 3 | 19
  5-19Y, MHCM, nets - not present: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM, nets - not present | 162 | 41 | 14 | 13 | 276
  5-19Y, MHCM, nets - present on all windows: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM, nets - present on all windows | 17 | 5 | 2 | 0 | 25
  5-19Y, MHCM, nets - present on some windows: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MHCM, nets - present on some windows | 19 | 5 | 0 | 0 | 27
  20+Y, MHCM roof - grass/palm: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM roof - grass/palm | 27 | 0 |  | 1 | 98
  20+Y, MHCM roof - iron sheet: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM roof - iron sheet | 56 | 4 |  | 0 | 394
  20+Y, MHCM roof - other: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM roof - other | 4 | 0 |  | 1 | 16
  20+Y, MHCM windows/eaves - closed: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM windows/eaves - closed | 64 | 4 |  | 1 | 421
  20+Y, MHCM windows/eaves - open: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM windows/eaves - open | 9 | 0 |  | 0 | 33
  20+Y, MHCM windows/eaves - partially open: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM windows/eaves - partially open | 14 | 0 |  | 0 | 54
  20+Y, MHCM, nets - not present: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM, nets - not present | 74 | 4 |  | 1 | 438
  20+Y, MHCM, nets - present on all windows: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM, nets - present on all windows | 7 | 0 |  | 0 | 32
  20+Y, MHCM, nets - present on some windows: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MHCM, nets - present on some windows | 6 | 0 |  | 0 | 38

44. Secondary Outcome: Number of Subjects Classified by House Information Regarding Main Source of the Drinking Water and Presence of Electricity at Survey 1
Description: The malaria prevention and risk factors characteristics were the following: Main source of drinking water (MSDW): bottled water, closed water source (piped water, tube well, dug well, protected well), open water source (unprotected well, spring water, rainwater, tanker truck, surface water), missing; and Presence of electricity (PE): Yes, No, missing.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 1) | Medium PD Group (Survey 1) | High PD Group (Survey 1) | Very High PD Group (Survey 1) | Neg PD Group (Survey 1)
Number analyzed (Participants) | 786 | 258 | 81 | 188 | 5088
Participants
  6M-4Y, MSDW - bottled water: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MSDW - bottled water | 1 | 0 | 0 | 0 | 22
  6M-4Y, MSDW - closed water source: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MSDW - closed water source | 246 | 111 | 28 | 49 | 1637
  6M-4Y, MSDW - open water source: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, MSDW - open water source | 126 | 59 | 30 | 70 | 821
  6M-4Y, PE - Yes: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PE - Yes | 66 | 24 | 7 | 13 | 780
  6M-4Y, PE - No: number analyzed (Participants) | 373 | 170 | 58 | 119 | 2480
  6M-4Y, PE - No | 307 | 146 | 51 | 106 | 1700
  5-19Y, MSDW - bottled water: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MSDW - bottled water | 1 | 0 | 0 | 0 | 9
  5-19Y, MSDW - closed water source: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MSDW - closed water source | 182 | 41 | 13 | 19 | 767
  5-19Y, MSDW - open water source: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MSDW - open water source | 111 | 30 | 10 | 39 | 390
  5-19Y, MSDW - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, MSDW - missing | 0 | 0 | 0 | 0 | 1
  5-19Y, PE - Yes: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PE - Yes | 48 | 13 | 4 | 4 | 384
  5-19Y, PE - No: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PE - No | 246 | 58 | 19 | 54 | 782
  5-19Y, PE - missing: number analyzed (Participants) | 294 | 71 | 23 | 58 | 1167
  5-19Y, PE - missing | 0 | 0 | 0 | 0 | 1
  20+Y, MSDW - bottled water: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MSDW - bottled water | 1 | 0 |  | 0 | 12
  20+Y, MSDW - closed water source: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MSDW - closed water source | 82 | 10 |  | 4 | 943
  20+Y, MSDW - open water source: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MSDW - open water source | 36 | 7 |  | 7 | 485
  20+Y, MSDW - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, MSDW - missing | 0 | 0 |  | 0 | 1
  20+Y, PE - Yes: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PE - Yes | 18 | 5 |  | 1 | 397
  20+Y, PE - No: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PE - No | 101 | 12 |  | 10 | 1043
  20+Y, PE - missing: number analyzed (Participants) | 119 | 17 | 0 | 11 | 1441
  20+Y, PE - missing | 0 | 0 |  | 0 | 1

45. Secondary Outcome: Number of Subjects Classified by House Information Regarding Main Source of the Drinking Water and Presence of Electricity at Survey 2
Description: The malaria prevention and risk factors characteristics were the following: Main source of drinking water (MSDW): bottled water, closed water source (piped water, tube well, dug well, protected well), open water source (unprotected well, spring water, rainwater, tanker truck, surface water); and Presence of electricity (PE): Yes, No.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 2) | Medium PD Group (Survey 2) | High PD Group (Survey 2) | Very High PD Group (Survey 2) | Neg PD Group (Survey 2)
Number analyzed (Participants) | 740 | 229 | 101 | 119 | 5222
Participants
  6M-4Y, MSDW - bottled water: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MSDW - bottled water | 1 | 0 | 0 | 0 | 4
  6M-4Y, MSDW - closed water source: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MSDW - closed water source | 207 | 93 | 44 | 42 | 1784
  6M-4Y, MSDW - open water source: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, MSDW - open water source | 75 | 55 | 23 | 34 | 835
  6M-4Y, PE - Yes: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PE - Yes | 49 | 18 | 9 | 9 | 824
  6M-4Y, PE - No: number analyzed (Participants) | 283 | 148 | 67 | 76 | 2623
  6M-4Y, PE - No | 234 | 130 | 58 | 67 | 1799
  5-19Y, MSDW - bottled water: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MSDW - bottled water | 1 | 0 | 0 | 0 | 3
  5-19Y, MSDW - closed water source: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MSDW - closed water source | 229 | 45 | 22 | 21 | 760
  5-19Y, MSDW - open water source: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, MSDW - open water source | 103 | 26 | 7 | 15 | 395
  5-19Y, PE - Yes: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PE - Yes | 60 | 12 | 11 | 4 | 366
  5-19Y, PE - No: number analyzed (Participants) | 333 | 71 | 29 | 36 | 1158
  5-19Y, PE - No | 273 | 59 | 18 | 32 | 792
  20+Y, MSDW - bottled water: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MSDW - bottled water | 0 | 0 | 0 | 0 | 4
  20+Y, MSDW - closed water source: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MSDW - closed water source | 87 | 7 | 4 | 1 | 987
  20+Y, MSDW - open water source: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, MSDW - open water source | 37 | 3 | 1 | 6 | 450
  20+Y, PE - Yes: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PE - Yes | 23 | 4 | 2 | 1 | 436
  20+Y, PE - No: number analyzed (Participants) | 124 | 10 | 5 | 7 | 1441
  20+Y, PE - No | 101 | 6 | 3 | 6 | 1005

46. Secondary Outcome: Number of Subjects Classified by House Information Regarding Main Source of the Drinking Water and Presence of Electricity at Survey 3
Description: The malaria prevention and risk factors characteristics were the following: Main source of drinking water (MSDW): bottled water, closed water source (piped water, tube well, dug well, protected well), open water source (unprotected well, spring water, rainwater, tanker truck, surface water); and Presence of electricity (PE): Yes, No.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 3) | Medium PD Group (Survey 3) | High PD Group (Survey 3) | Very High PD Group (Survey 3) | Neg PD Group (Survey 3)
Number analyzed (Participants) | 791 | 268 | 92 | 130 | 5119
Participants
  6M-4Y, MSDW - bottled water: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MSDW - bottled water | 0 | 0 | 0 | 1 | 26
  6M-4Y, MSDW - closed water source: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MSDW - closed water source | 185 | 97 | 37 | 53 | 1613
  6M-4Y, MSDW - open water source: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, MSDW - open water source | 94 | 64 | 37 | 37 | 949
  6M-4Y, PE - Yes: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PE - Yes | 36 | 25 | 8 | 11 | 775
  6M-4Y, PE - No: number analyzed (Participants) | 279 | 161 | 74 | 91 | 2588
  6M-4Y, PE - No | 243 | 136 | 66 | 80 | 1813
  5-19Y, MSDW - bottled water: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MSDW - bottled water | 0 | 1 | 0 | 0 | 13
  5-19Y, MSDW - closed water source: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MSDW - closed water source | 214 | 51 | 6 | 23 | 715
  5-19Y, MSDW - open water source: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, MSDW - open water source | 127 | 42 | 7 | 12 | 401
  5-19Y, PE - Yes: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PE - Yes | 56 | 19 | 5 | 7 | 348
  5-19Y, PE - No: number analyzed (Participants) | 341 | 94 | 13 | 35 | 1129
  5-19Y, PE - No | 285 | 75 | 8 | 28 | 781
  20+Y, MSDW - bottled water: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MSDW - bottled water | 0 | 0 | 0 | 0 | 15
  20+Y, MSDW - closed water source: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MSDW - closed water source | 101 | 8 | 2 | 1 | 884
  20+Y, MSDW - open water source: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, MSDW - open water source | 70 | 5 | 3 | 3 | 503
  20+Y, PE - Yes: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PE - Yes | 19 | 3 | 0 | 1 | 386
  20+Y, PE - No: number analyzed (Participants) | 171 | 13 | 5 | 4 | 1402
  20+Y, PE - No | 152 | 10 | 5 | 3 | 1016

47. Secondary Outcome: Number of Subjects Classified by House Information Regarding Main Source of the Drinking Water and Presence of Electricity at Survey 4
Description: The malaria prevention and risk factors characteristics were the following: Main source of drinking water (MSDW): bottled water, closed water source (piped water, tube well, dug well, protected well), open water source (unprotected well, spring water, rainwater, tanker truck, surface water); and Presence of electricity (PE): Yes, No.
  Data were collected across centers from subjects between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4. Results were presented per the following P. falciparum parasite density status subgroups: Low, Medium, High, Very high, and Negative (Neg).
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group (Survey 4) | Medium PD Group (Survey 4) | High PD Group (Survey 4) | Very High PD Group (Survey 4) | Neg PD Group (Survey 4)
Number analyzed (Participants) | 453 | 158 | 36 | 68 | 1684
Participants
  6M-4Y, MSDW - bottled water: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MSDW - bottled water | 0 | 0 | 0 | 0 | 1
  6M-4Y, MSDW - closed water source: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MSDW - closed water source | 139 | 79 | 15 | 38 | 656
  6M-4Y, MSDW - open water source: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, MSDW - open water source | 29 | 24 | 5 | 16 | 191
  6M-4Y, PE - Yes: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, PE - Yes | 20 | 5 | 0 | 3 | 384
  6M-4Y, PE - No: number analyzed (Participants) | 168 | 107 | 20 | 54 | 848
  6M-4Y, PE - No | 148 | 98 | 20 | 51 | 464
  5-19Y, MSDW - bottled water: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MSDW - bottled water | 0 | 0 | 0 | 0 | 0
  5-19Y, MSDW - closed water source: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MSDW - closed water source | 155 | 38 | 12 | 9 | 247
  5-19Y, MSDW - open water source: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, MSDW - open water source | 43 | 13 | 4 | 4 | 81
  5-19Y, PE - Yes: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PE - Yes | 23 | 8 | 3 | 4 | 161
  5-19Y, PE - No: number analyzed (Participants) | 198 | 51 | 16 | 13 | 328
  5-19Y, PE - No | 175 | 43 | 13 | 9 | 167
  20+Y, MSDW - bottled water: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MSDW - bottled water | 0 | 0 |  | 0 | 1
  20+Y, MSDW - closed water source: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MSDW - closed water source | 69 | 2 |  | 1 | 391
  20+Y, MSDW - open water source: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, MSDW - open water source | 18 | 2 |  | 0 | 116
  20+Y, PE - Yes: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PE - Yes | 9 | 2 |  | 0 | 206
  20+Y, PE - No: number analyzed (Participants) | 87 | 4 | 0 | 1 | 508
  20+Y, PE - No | 78 | 2 |  | 1 | 302

48. Secondary Outcome: Number of Subjects With Malaria Prevention Measures (MPM) at Each Survey
Description: The malaria prevention measures (MPM) data were collected across centers from subjects with age between and including: 6M-4Y, 5-19 Y and 20Y+, for each Survey.
  The MPM results include the following categories: Use of Mosquito coils over 7 days (UMc > 7D), Use of Insecticide spray over 7 days (UIs > 7D), Use of Commercial Repellents over 7 days (UCR > 7D), Use of Traditional Repellents over 7 days (UTR > 7D), Use of none of above over 7 days (Una >7D), Use of indoor residual spray in past 12 months to spray interior walls (Uirs past 12M), Use of indoor residual spray - number of months ago (Uirs-nM) or Use of indoor residual spray- no spray (Uirs-no spray): the number of months ago for each Uirs-nM sub-categories is defined using the following [x Months]. Not all Uirs-nM sub-categories were analyzed in each survey.
Time Frame: At each Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Number analyzed (Participants) | 6401 | 6411 | 6400 | 2399
Participants
  [6M-4Y], UMc > 7D, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UMc > 7D, Yes | 433 | 398 | 348 | 239
  [6M-4Y], UMc > 7D, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UMc > 7D, Missing/No | 2767 | 2799 | 2845 | 954
  [6M-4Y], UIs > 7D, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UIs > 7D, Yes | 101 | 60 | 48 | 27
  [6M-4Y], UIs > 7D, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UIs > 7D, Missing/No | 3099 | 3137 | 3145 | 1166
  [6M-4Y], UCR > 7D, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UCR > 7D, Yes | 4 | 5 | 24 | 20
  [6M-4Y], UCR > 7D, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UCR > 7D, Missing/No | 3196 | 3192 | 3169 | 1173
  [6M-4Y], UTR > 7D, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UTR > 7D, Yes | 7 | 9 | 0 | 2
  [6M-4Y], UTR > 7D, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], UTR > 7D, Missing/No | 3193 | 3188 | 3193 | 1191
  [6M-4Y], Una >7D, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Una >7D, Yes | 2663 | 2726 | 2778 | 905
  [6M-4Y], Una >7D, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Una >7D, Missing/No | 537 | 471 | 415 | 288
  [6M-4Y], Uirs past 12M, Yes: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Uirs past 12M, Yes | 59 | 15 | 7 | 3
  [6M-4Y], Uirs past 12M, Missing/No: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Uirs past 12M, Missing/No | 3141 | 3182 | 3186 | 1190
  [6M-4Y], Uirs-nM [1 Month]: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Uirs-nM [1 Month] | 9 | 1 | 1 | 0
  [6M-4Y], Uirs-nM [11 Months]: number analyzed (Participants) | 0 | 0 | 3193 | 0
  [6M-4Y], Uirs-nM [11 Months] |  |  | 1 |
  [6M-4Y], Uirs-nM [12 Months]: number analyzed (Participants) | 3200 | 3197 | 3193 | 0
  [6M-4Y], Uirs-nM [12 Months] | 5 | 1 | 2 |
  [6M-4Y], Uirs-nM [10 Months]: number analyzed (Participants) | 0 | 0 | 0 | 1193
  [6M-4Y], Uirs-nM [10 Months] |  |  |  | 1
  [6M-4Y], Uirs-nM [2 Months]: number analyzed (Participants) | 3200 | 3197 | 0 | 1193
  [6M-4Y], Uirs-nM [2 Months] | 6 | 3 |  | 1
  [6M-4Y], Uirs-nM [3 Months]: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Uirs-nM [3 Months] | 21 | 5 | 3 | 1
  [6M-4Y], Uirs-nM [4 Months]: number analyzed (Participants) | 3200 | 3197 | 3193 | 0
  [6M-4Y], Uirs-nM [4 Months] | 9 | 2 | 1 |
  [6M-4Y], Uirs-nM [5 Months]: number analyzed (Participants) | 3200 | 3197 | 0 | 0
  [6M-4Y], Uirs-nM [5 Months] | 1 | 2 |  |
  [6M-4Y], Uirs-nM [6 Months]: number analyzed (Participants) | 3200 | 0 | 0 | 0
  [6M-4Y], Uirs-nM [6 Months] | 6 |  |  |
  [6M-4Y], Uirs-nM [7 Months]: number analyzed (Participants) | 3200 | 3197 | 0 | 0
  [6M-4Y], Uirs-nM [7 Months] | 1 | 1 |  |
  [6M-4Y], Uirs-nM [9 Months]: number analyzed (Participants) | 3200 | 0 | 0 | 0
  [6M-4Y], Uirs-nM [9 Months] | 1 |  |  |
  [6M-4Y], Uirs-nM [no spray]: number analyzed (Participants) | 3200 | 3197 | 3193 | 1193
  [6M-4Y], Uirs-nM [no spray] | 3141 | 3182 | 3186 | 1190
  [5-19Y], UMc > 7D, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UMc > 7D, Yes | 227 | 209 | 180 | 127
  [5-19Y], UMc > 7D, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UMc > 7D, Missing/No | 1386 | 1418 | 1432 | 479
  [5-19Y], UIs > 7D, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UIs > 7D, Yes | 45 | 32 | 20 | 10
  [5-19Y], UIs > 7D, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UIs > 7D, Missing/No | 1568 | 1595 | 1592 | 596
  [5-19Y], UCR > 7D, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UCR > 7D, Yes | 4 | 2 | 12 | 7
  [5-19Y], UCR > 7D, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UCR > 7D, Missing/No | 1609 | 1625 | 1600 | 599
  [5-19Y], UTR > 7D, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UTR > 7D, Yes | 3 | 3 | 0 | 2
  [5-19Y], UTR > 7D, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], UTR > 7D, Missing/No | 1610 | 1624 | 1612 | 604
  [5-19Y], Una >7D, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Una >7D, Yes | 1336 | 1381 | 1401 | 460
  [5-19Y], Una >7D, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Una >7D, Missing/No | 277 | 246 | 211 | 146
  [5-19Y], Uirs past 12M, Yes: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Uirs past 12M, Yes | 24 | 8 | 3 | 1
  [5-19Y], Uirs past 12M, Missing/No: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Uirs past 12M, Missing/No | 1589 | 1619 | 1609 | 605
  [5-19Y], Uirs-nM [1 Month]: number analyzed (Participants) | 1613 | 1627 | 0 | 606
  [5-19Y], Uirs-nM [1 Month] | 2 | 1 |  | 1
  [5-19Y], Uirs-nM [11 Months]: number analyzed (Participants) | 0 | 0 | 1612 | 0
  [5-19Y], Uirs-nM [11 Months] |  |  | 1 |
  [5-19Y], Uirs-nM [12 Months]: number analyzed (Participants) | 1613 | 1627 | 1612 | 0
  [5-19Y], Uirs-nM [12 Months] | 2 | 1 | 1 |
  [5-19Y], Uirs-nM [10 Months]: number analyzed (Participants) | 0 | 0 | 0 | 0
  [5-19Y], Uirs-nM [2 Months]: number analyzed (Participants) | 1613 | 1627 | 0 | 606
  [5-19Y], Uirs-nM [2 Months] | 1 | 2 |  | 0
  [5-19Y], Uirs-nM [3 Months]: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Uirs-nM [3 Months] | 13 | 3 | 0 | 0
  [5-19Y], Uirs-nM [4 Months]: number analyzed (Participants) | 1613 | 1627 | 1612 | 0
  [5-19Y], Uirs-nM [4 Months] | 2 | 0 | 1 |
  [5-19Y], Uirs-nM [5 Months]: number analyzed (Participants) | 1613 | 1627 | 0 | 0
  [5-19Y], Uirs-nM [5 Months] | 0 | 1 |  |
  [5-19Y], Uirs-nM [6 Months]: number analyzed (Participants) | 1613 | 0 | 0 | 0
  [5-19Y], Uirs-nM [6 Months] | 4 |  |  |
  [5-19Y], Uirs-nM [7 Months]: number analyzed (Participants) | 1613 | 1627 | 0 | 0
  [5-19Y], Uirs-nM [7 Months] | 0 | 0 |  |
  [5-19Y], Uirs-nM [9 Months]: number analyzed (Participants) | 1613 | 0 | 0 | 0
  [5-19Y], Uirs-nM [9 Months] | 0 |  |  |
  [5-19Y], Uirs-nM [no spray]: number analyzed (Participants) | 1613 | 1627 | 1612 | 606
  [5-19Y], Uirs-nM [no spray] | 1589 | 1619 | 1609 | 605
  [Y20+], UMc > 7D, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UMc > 7D, Yes | 196 | 199 | 167 | 117
  [Y20+], UMc > 7D, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UMc > 7D, Missing/No | 1392 | 1388 | 1428 | 483
  [Y20+], UIs > 7D, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UIs > 7D, Yes | 46 | 30 | 28 | 11
  [Y20+], UIs > 7D, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UIs > 7D, Missing/No | 1542 | 1557 | 1567 | 589
  [Y20+], UCR > 7D, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UCR > 7D, Yes | 0 | 4 | 12 | 12
  [Y20+], UCR > 7D, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UCR > 7D, Missing/No | 1588 | 1583 | 1583 | 588
  [Y20+], UTR > 7D, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UTR > 7D, Yes | 4 | 4 | 0 | 0
  [Y20+], UTR > 7D, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], UTR > 7D, Missing/No | 1584 | 1583 | 1595 | 600
  [Y20+], Una >7D, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Una >7D, Yes | 1346 | 1350 | 1392 | 460
  [Y20+], Una >7D, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Una >7D, Missing/No | 242 | 237 | 203 | 140
  [Y20+], Uirs past 12M, Yes: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Uirs past 12M, Yes | 32 | 7 | 2 | 2
  [Y20+], Uirs past 12M, Missing/No: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Uirs past 12M, Missing/No | 1556 | 1580 | 1593 | 598
  [Y20+], Uirs-nM [1 Month]: number analyzed (Participants) | 1588 | 1587 | 0 | 600
  [Y20+], Uirs-nM [1 Month] | 7 | 0 |  | 0
  [Y20+], Uirs-nM [11 Months]: number analyzed (Participants) | 0 | 0 | 1595 | 0
  [Y20+], Uirs-nM [11 Months] |  |  | 0 |
  [Y20+], Uirs-nM [12 Months]: number analyzed (Participants) | 1588 | 1587 | 1595 | 0
  [Y20+], Uirs-nM [12 Months] | 3 | 0 | 1 |
  [Y20+], Uirs-nM [10 Months]: number analyzed (Participants) | 0 | 0 | 0 | 600
  [Y20+], Uirs-nM [10 Months] |  |  |  | 1
  [Y20+], Uirs-nM [2 Months]: number analyzed (Participants) | 1588 | 1587 | 0 | 600
  [Y20+], Uirs-nM [2 Months] | 4 | 1 |  | 1
  [Y20+], Uirs-nM [3 Months]: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Uirs-nM [3 Months] | 8 | 3 | 1 | 0
  [Y20+], Uirs-nM [4 Months]: number analyzed (Participants) | 1588 | 1587 | 1595 | 0
  [Y20+], Uirs-nM [4 Months] | 6 | 2 | 0 |
  [Y20+], Uirs-nM [5 Months]: number analyzed (Participants) | 1588 | 1587 | 0 | 0
  [Y20+], Uirs-nM [5 Months] | 1 | 1 |  |
  [Y20+], Uirs-nM [6 Months]: number analyzed (Participants) | 1588 | 0 | 0 | 0
  [Y20+], Uirs-nM [6 Months] | 2 |  |  |
  [Y20+], Uirs-nM [7 Months]: number analyzed (Participants) | 1588 | 1587 | 0 | 0
  [Y20+], Uirs-nM [7 Months] | 1 | 0 |  |
  [Y20+], Uirs-nM [9 Months]: number analyzed (Participants) | 1588 | 0 | 0 | 0
  [Y20+], Uirs-nM [9 Months] | 0 |  |  |
  [Y20+], Uirs-nM [no spray]: number analyzed (Participants) | 1588 | 1587 | 1595 | 600
  [Y20+], Uirs-nM [no spray] | 1556 | 1580 | 1593 | 598

49. Secondary Outcome: Number of Subjects With Plasmodium Species Other Than P. Falciparum at Survey 1
Description: Data were collected across centers from subjects with age between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 1.
  The other Plasmodium species assessed were: P. Malaria, P. Vivax, P. Ovale. Infection were determined using a blood smear slide, and categorized according positive (Pos) and negative (Neg) results.
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Group (6M-4Y) (Survey 1): Subjects from Survey 1, aged between and including 6 months (6M) to 4 years (4Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (5-19Y) (Survey 1): Subjects from Survey 1, aged 5 to 19 years (5-19Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (20Y+) (Survey 1): Subjects from Survey 1, aged 20 years or older (20Y+), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
Arm/Group | Overall Study Group (6M-4Y) (Survey 1) | Overall Study Group (5-19Y) (Survey 1) | Overall Study Group (20Y+) (Survey 1)
Number analyzed (Participants) | 3200 | 1613 | 1588
Participants
  P.Malariae, Pos | 19 | 21 | 1
  P.Malariae, Neg | 3181 | 1592 | 1587
  P.Vivax, Pos | 0 | 0 | 0
  P.Vivax, Neg | 3200 | 1613 | 1588
  P.Ovale, Pos | 3 | 1 | 0
  P.Ovale, Neg | 3197 | 1612 | 1588

50. Secondary Outcome: Number of Subjects With Plasmodium Species Other Than P. Falciparum at Survey 2
Description: Data were collected across centers from subjects with age between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 2.
  The other Plasmodium species assessed were: P. Malaria, P. Vivax, P. Ovale. Infection were determined using a blood smear slide, and categorized according positive (Pos) and negative (Neg) results.
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Group (6M-4Y) (Survey 2): Subjects from Survey 2, aged between and including 6 months (6M) to 4 years (4Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (5-19Y) (Survey 2): Subjects from Survey 2, aged 5 to 19 years (5-19Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (20Y+) (Survey 2): Subjects from Survey 2, aged 20 years or older (20Y+), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
Arm/Group | Overall Study Group (6M-4Y) (Survey 2) | Overall Study Group (5-19Y) (Survey 2) | Overall Study Group (20Y+) (Survey 2)
Number analyzed (Participants) | 3197 | 1627 | 1587
Participants
  P.Malariae, Pos | 32 | 27 | 2
  P.Malariae, Neg | 3165 | 1600 | 1585
  P.Vivax, Pos | 0 | 0 | 0
  P.Vivax, Neg | 3197 | 1627 | 1587
  P.Ovale, Pos | 6 | 3 | 2
  P.Ovale, Neg | 3191 | 1624 | 1585

51. Secondary Outcome: Number of Subjects With Plasmodium Species Other Than P. Falciparum at Survey 3
Description: Data were collected across centers from subjects with age between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 3.
  The other Plasmodium species assessed were: P. Malaria, P. Vivax, P. Ovale. Infection were determined using a blood smear slide, and categorized according positive (Pos) and negative (Neg) results.
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Group (6M-4Y) (Survey 3): Subjects from Survey 3, aged between and including 6 months (6M) to 4 years (4Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (5-19Y) (Survey 3): Subjects from Survey 3, aged 5 to 19 years (5-19Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (20Y+) (Survey 3): Subjects from Survey 3, aged 20 years or older (20Y+), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
Arm/Group | Overall Study Group (6M-4Y) (Survey 3) | Overall Study Group (5-19Y) (Survey 3) | Overall Study Group (20Y+) (Survey 3)
Number analyzed (Participants) | 3193 | 1612 | 1595
Participants
  P.Malariae, Pos | 48 | 27 | 0
  P.Malariae, Neg | 3145 | 1585 | 1595
  P.Vivax, Pos | 0 | 0 | 0
  P.Vivax, Neg | 3193 | 1612 | 1595
  P.Ovale, Pos | 6 | 4 | 1
  P.Ovale, Neg | 3187 | 1608 | 1594

52. Secondary Outcome: Number of Subjects With Plasmodium Species Other Than P. Falciparum at Survey 4
Description: Data were collected across centers from subjects with age between and including: 6M-4Y, 5-19 Y and 20Y+, for Survey 4.
  The other Plasmodium species assessed were: P. Malaria, P. Vivax, P. Ovale. Infection were determined using a blood smear slide, and categorized according positive (Pos) and negative (Neg) results.
Time Frame: At Survey visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Group (6M-4Y) (Survey 4): Subjects from Survey 4, aged between and including 6 months (6M) to 4 years (4Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (5-19Y) (Survey 4): Subjects from Survey 4, aged 5 to 19 years (5-19Y), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
- Overall Study Group (20Y+) (Survey 4): Subjects from Survey 4, aged 20 years or older (20Y+), enrolled in catchment areas of study 110021 (NCT00866619), infected with P. falciparum parasite. Infection determined using a blood smear slide and determined using microscopy.
Arm/Group | Overall Study Group (6M-4Y) (Survey 4) | Overall Study Group (5-19Y) (Survey 4) | Overall Study Group (20Y+) (Survey 4)
Number analyzed (Participants) | 1193 | 606 | 600
Participants
  P.Malariae, Pos | 32 | 28 | 0
  P.Malariae, Neg | 1161 | 578 | 600
  P.Vivax, Pos | 0 | 0 | 0
  P.Vivax, Neg | 1193 | 606 | 600
  P.Ovale, Pos | 3 | 3 | 1
  P.Ovale, Neg | 1190 | 603 | 599

53. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to Study Procedure for Each Survey
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Capillary blood sampling was the only invasive procedure involved in this study. SAEs related to this procedure were recorded at the Survey visit.
Time Frame: At each Survey visit
Population: The analysis was performed on the Total cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
Number analyzed (Participants) | 6404 | 6414 | 6400 | 2400
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Capillary blood sampling was the only invasive procedure involved in this study. Serious adverse events (SAEs) related to this procedure were recorded at each survey visit.
Description: Anticipated and unanticipated adverse events symptoms were not collected in the study.
Arm/Group | Overall Study Group (Survey 1) | Overall Study Group (Survey 2) | Overall Study Group (Survey 3) | Overall Study Group (Survey 4)
All-Cause Mortality (participants affected / at risk) | 0/6404 | 0/6414 | 0/6400 | 0/2400
Serious Adverse Events (participants affected / at risk) | 0/6404 | 0/6414 | 0/6400 | 0/2400
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.